CLINICAL TRIAL: NCT04585815
Title: A Phase 1b/2 Open Label Umbrella Study of Sasanlimab Combined With Anti-Cancer Therapies Targeting Multiple Molecular Mechanisms in Participants With Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study of Immunotherapy (Sasanlimab) in Combination With Targeted Therapies in People With Advanced Non-small Cell Lung Cancer (NSCLC) (Landscape 1011 Study)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to portfolio re-prioritization and strategic considerations. The decision was not based on any safety concerns and/or regulatory interactions
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B8011011; 2020-002829-28 (EudraCT Number)
Record Dates: First submitted 2020-09-30; First posted 2020-10-14 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-Small-Cell Lung Carcinoma; NSCLC; non small cell lung cancer; non-small cell lung cancer; BRAF mutation; BRAF V600e; BRAF; B-RAF NSCLC; lung cancer; immunotherapy; sasanlimab; encorafenib; binimetinib; axitinib; SEA-TGT; TIGIT; locally advanced; metastatic; ECOG 0; ECOG 1; Stage 3B; Stage IV; previously untreated; second-line therapy; first-line therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasm Metastasis | interventions — encorafenib; binimetinib; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sub-Study A (Experimental): Sasanlimab will be administered subcutaneously. Encorafenib & binimetinib will be administered orally. Treatments will be administered until progressive disease, unacceptable AE, participant withdraws, or study is terminated.
  Interventions: Drug: Sasanlimab Prefilled syringe; Drug: Encorafenib; Drug: Binimetinib
- Sub-Study B (Experimental): Sasanlimab will be administered subcutaneously. Axitinib will be administered orally. SEA-TGT will be administered intravenously. Treatments will be administered until progressive disease, unacceptable AE, patient withdraws, or study is terminated.
  Interventions: Drug: Sasanlimab; Drug: Axitinib; Drug: SEA-TGT

INTERVENTIONS:
Drug: Sasanlimab Prefilled syringe — prefilled syringe
  Arms: Sub-Study A
Drug: Encorafenib — capsules
  Arms: Sub-Study A
Drug: Binimetinib — tablets
  Arms: Sub-Study A
Drug: Sasanlimab — solution supplied in vials
  Arms: Sub-Study B
Drug: Axitinib — tablets
  Arms: Sub-Study B
Drug: SEA-TGT — solution in vials
  Arms: Sub-Study B

SUMMARY:
Phase 1b/Phase 2 Umbrella Study; open-label, multi-center, parallel group study.

Sasanlimab (a PD-1 antagonist monoclonal antibody) will be combined with a different targeted therapy in each sub-study. Phase1b of each sub-study will evaluate the safety of the combination and select the dose for the Phase 2 portion. Phase 2 of each sub-study will evaluate the anti-tumor activity of the combination.

Sub-Study A is active, not recruiting, ongoing participants are still receiving treatment in Phase 1, Phase 2 will not be initiated.

Sub-study B is complete. All participants have discontinued treatment and any additional follow up required by protocol.

DETAILED DESCRIPTION:
Landscape 1011 is a clinical research study for people with advanced (stage 3b or 4) non-small cell lung cancer (NSCLC). The purpose of this study is to learn if the study medicine (sasanlimab, a type of immunotherapy) along with other study medicines is safe and effective in people with non-small cell lung cancer that has spread outside of the lungs. There are currently two sub-studies using different types of medicines. People in the first sub-study will receive sasanlimab as a subcutaneous (under the skin) injection at the study clinic every 4 weeks. Additionally, they will take targeted cancer therapies encorafenib by mouth once a day and binimetinib by mouth twice a day at home.

People in the second sub-study will receive the study medicine sasanlimab as a subcutaneous (under the skin) injection at the study clinic every 3 weeks and will also receive SEA-TGT (an immunotherapy) by infusion every three weeks.

Additionally, they will take axitinib (a targeted therapy) by mouth twice a day at home.

In addition to taking the study drugs, participants in the sub-studies will be asked to visit the clinic for health checks. These include health questions, physical examinations, blood and urine samples, and imaging scans. These assessments help the study doctor and team to monitor the participants' safety and well-being, and to see how their cancer is responding to the treatment. Participants will continue in the study until the cancer is no longer responding to the study medicine.

ELIGIBILITY:
Inclusion Criteria Umbrella Phase 1b & 2:

* Histologically or cytologically confirmed locally advanced/metastatic (Stage IIIB-IV) NSCLC.
* At least one measurable lesion per RECIST v1.1 at Screening.
* ECOG Performance Status 0 or 1.
* Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade ≤1.
* Adequate hepatic, renal, and bone marrow function.

Additional Inclusion Criteria for Sub-Study A Phase 1b &2:

-BRAFV600E mutation in tumor tissue or plasma as determined by a local laboratory PCR or NGS assay and documented in a local pathology report.

Additional Inclusion Criteria for Sub-Study A Phase 1b only:

-Any line of therapy for locally advanced/metastatic NSCLC.

Additional Inclusion Criteria for Sub-Study A Phase 2 only:

-Previously untreated for locally advanced/metastatic NSCLC

Additional Inclusion Criteria for Sub-Study B Phase 1b only::

-Any line of therapy for locally advanced/metastatic NSCLC.

Additional Inclusion Criteria for Sub-Study B Phase 2 only:

* Previously untreated for locally advanced/metastatic NSCLC (Arms B1 & B2), or
* One or 2 prior lines of therapy for advanced/metastatic NSCLC (Arm B3), including immune checkpoint inhibitor treatment + chemotherapy, and have progressed during or after that therapy.
* PD-L1 TPS ≥1%

Exclusion Criteria Umbrella Phase 1b &2:

* Active or prior autoimmune disease that might deteriorate when receiving an immunostimulatory agent.
* Active non-infectious pneumonitis, pulmonary fibrosis, or known history of immune-mediated pneumonitis.
* Active infection requiring systemic therapy.
* Clinically significant cardiovascular disease.
* Other malignancy within 2 years of first dose, with exceptions.
* Symptomatic brain metastasis, with exceptions.

Additional Exclusion Criteria for Sub-Study A Phase 1b&2:

* EGFR mutation, ALK fusion oncogene, or ROS1 rearrangement.
* Prior treatment with any BRAF inhibitor or MEK inhibitor.

Additional Exclusion Criteria for Sub-Study A Phase 2 only:

-Prior therapy with anti-PD-1, anti-PD-L1, or anti-PD-L2 agents.

Additional Exclusion Criteria for Sub-Study B Phase 1b&2:

-Documentation of any tumor-driving molecular alteration (eg, BRAF, EGFR, ALK)

Additional Exclusion Criteria for Sub-Study B Phase 2 only:

* Prior therapy with anti-PD-1, anti-PD-L1, or anti-PD-L2 agents.(Arms B1 & B2)
* Confirmed progressive disease on 1st or 2nd imaging tumor assessment after initiation of therapy for advanced/metastatic NSCLC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2024-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (51):
- United States (40):
  - City of Hope Investigational Drug Services (IDS), Duarte, California
  - City of Hope, Duarte, California
  - UCSD Medical Center - Encinitas, Encinitas, California
  - California Cancer Associates for Research and Excellence, Inc (cCARE), Fresno, California
  - The Oncology Institute of Hope and Innovation, Glendale, California
  - Koman Family Outpatient Pavilion, La Jolla, California
  - Sulpizio Cardiovascular Center at UC San Diego Health, La Jolla, California
  - UC San Diego Medical Center - La Jolla (Jacobs Medical Center / Thornton Pavilion), La Jolla, California
  - UC San Diego Moores Cancer Center - Investigational Drug Services, La Jolla, California
  - UCSD Perlman Medical Offices, La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - The Oncology Institute of Hope and Innovation, Long Beach, California
  - The Oncology Institute of Hope and Innovation, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - The Oncology Institute of Hope and Innovation, Santa Ana, California
  - UCSD Medical Center - Vista, Vista, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - AdventHealth Celebration Infusion Center, Celebration, Florida
  - AdventHealth Medical Group Oncology Research at Celebration, Celebration, Florida
  - Advent Health Orlando - Investigational Drug Services, Orlando, Florida
  - AdventHealth Orlando Infusion Center, Orlando, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Henry Ford Medical Center - Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Medical Center - Columbus, Novi, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Mount Sinai Hospital Pharmacy, New York, New York
  - Tennessee Oncology PLLC, Dickson, Tennessee
  - Tennessee Oncology PLLC, Franklin, Tennessee
  - Tennessee Oncology PLLC, Gallatin, Tennessee
  - Tennessee Oncology PLLC, Hendersonville, Tennessee
  - Tennessee Oncology PLLC, Hermitage, Tennessee
  - Tennessee Oncology PLLC, Lebanon, Tennessee
  - Tennessee Oncology PLLC, Murfreesboro, Tennessee
  - Sarah Cannon Research Institute - Pharmacy, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Tennessee Oncology PLLC, Shelbyville, Tennessee
  - Tennessee Oncology PLLC, Smyrna, Tennessee
- Australia (5):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Concord Hospital, Concord, New South Wales
  - GenesisCare North Shore, St Leonards, New South Wales
  - North Shore Radiology and Nuclear Medicine, St Leonards, New South Wales
  - Austin Health, Heidelberg, Victoria
- Belgium (2):
  - Antwerp University Hospital, Edegem, Antwerpen
  - UZ Leuven, Leuven
- Taiwan (4):
  - Chung Shan Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Koo Foundation Sun Yat -Sen Cancer Center, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B8011011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sub-study A (SSA) was planned to be conducted in 2 parts: Phase 1b and Phase 2. Due to a business decision, Phase 2 was not initiated, hence no participants were enrolled for Phase 2 of SSA. Sub-study B (SSB) was conducted in 2 parts: Phase 1b and Phase 2.
Pre-assignment Details: 57 participants signed informed consent and 34 participants were enrolled in the study. Of these 34 participants, 13 were enrolled in Sub-study A and 21 in Sub-study B (9 in Phase [Ph] 1b and 12 in Phase 2).
Groups:
- Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg): Participants with non-small cell lung cancer (NSCLC) with BRAFV600 mutations were administered a single dose of sasanlimab 300 milligrams (mg) subcutaneously on Day 1 of each cycle along with once daily (QD) oral dose of 300 mg encorafenib and twice daily (BID) oral dose of 45 mg binimetinib during each 28-day cycle.
- Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg): Participants with NSCLC with BRAFV600 mutations were administered a single dose of sasanlimab 300 mg subcutaneously on Day 1 of each cycle along with QD oral dose of 450 mg encorafenib and BID oral dose of 45 mg binimetinib during each 28-day cycle.
- Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg): Participants with NSCLC and who received any line of therapy for advanced/metastatic NSCLC were administered a single dose of sasanlimab 225 mg every 3 weeks (Q3W) subcutaneously along with BID oral dose of 5 mg axitinib on Day 1 of each cycle during each 21-day cycle.
- Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg): Participants with NSCLC and who received any line of therapy for advanced/metastatic NSCLC were administered a single dose of sasanlimab 225 mg Q3W subcutaneously along with BID oral dose of 5 mg axitinib on Day 1 of each cycle and Q3W intravenous (IV) infusion of 1 milligram per kilogram (mg/kg) SEA-TGT on Day 1 of each cycle during each 21-day cycle.
- Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg): Participants with NSCLC with who were treatment-naïve for advanced/metastatic disease with low programmed death ligand - 1 (PD-L1) levels Tumor proportion score (TPS)-49 percent (%) were administered a single dose of sasanlimab 225 mg Q3W subcutaneously along with BID oral dose of 5 mg axitinib on Day 1 of each cycle and Q3W IV infusion of 1 mg/kg SEA-TGT on Day 1 of each cycle during each 21-day cycle.
- Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg): Participants with NSCLC with who were treatment-naïve for advanced/metastatic disease with high PD-L1 (TPS greater than or equal to [>=]50%) were administered a single dose of sasanlimab 225 mg Q3W subcutaneously along with BID oral dose of 5 mg axitinib on Day 1 of each cycle and Q3W IV infusion of 1 mg/kg SEA+ TGT on Day 1 of each cycle during each 21-day cycle.
- Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg): Participants with NSCLC who received 1 or 2 lines of therapy for advanced/metastatic NSCLC and whose disease has progressed on prior PD-1/ PD-L1 therapy and who have PD-L1 TPS >= 1% were administered a single dose of sasanlimab 225 mg Q3W subcutaneously along with BID oral dose of 5 mg axitinib on Day 1 of each cycle and 1 mg/kg IV infusion Q3W SEA-TGT on Day 1 of each cycle during each 21-day cycle.
Period: Sub-study A- Treatment Phase
Arm/Group | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg) | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg) | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
Started | 4 | 9 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 9 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Global deterioration of health status | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Sub-study A- Follow-up Phase
Arm/Group | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg) | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg) | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
Started | 2 (Eligible participants entered follow-up period following discontinuation of study treatment.) | 5 (Eligible participants entered follow-up period following discontinuation of study treatment.) | 0 | 0 | 0 | 0 | 0
Completed | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 1 | 3 | 0 | 0 | 0 | 0 | 0
Period: Sub-study B- Treatment Phase
Arm/Group | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg) | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg) | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
Started | 0 | 0 | 3 | 6 | 3 | 2 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 3 | 6 | 3 | 2 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 3 | 2 | 2 | 1 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Global deterioration of health status | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 1 | 0 | 0
Period: Sub-study B- Follow-up Phase
Arm/Group | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg) | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg) | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
Started | 0 | 0 | 2 (Eligible participants entered follow-up period following discontinuation of study treatment.) | 3 (Eligible participants entered follow-up period following discontinuation of study treatment.) | 3 (Eligible participants entered follow-up period following discontinuation of study treatment.) | 2 (Eligible participants entered follow-up period following discontinuation of study treatment.) | 6 (Eligible participants entered follow-up period following discontinuation of study treatment.)
Completed | 0 | 0 | 1 | 0 | 2 | 1 | 3
Not Completed | 0 | 0 | 1 | 3 | 1 | 1 | 3
Not completed — Death | 0 | 0 | 1 | 3 | 1 | 0 | 3
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who received at least 1 dose of study drug. Participants were classified according to the treatment actually received.
Groups:
- Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg): Participants with NSCLC with BRAFV600 mutations were administered a single dose of sasanlimab 300 mg subcutaneously on Day 1 of each cycle along with QD oral dose of 300 mg encorafenib and BID oral dose of 45 mg binimetinib during each 28-day cycle.
- Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg): Participants with NSCLC and who received any line of therapy for advanced/metastatic NSCLC were administered a single dose of sasanlimab 225 mg Q3W subcutaneously along with BID oral dose of 5 mg axitinib on Day 1 of each cycle during each 21-day cycle.
- Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg): Participants with NSCLC and who received any line of therapy for advanced/metastatic NSCLC were administered a single dose of sasanlimab 225 mg Q3W subcutaneously along with BID oral dose of 5 mg axitinib on Day 1 of each cycle and Q3W IV infusion of 1 mg/kg SEA-TGT on Day 1 of each cycle during each 21-day cycle.
- Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg): Participants with NSCLC with who were treatment-naïve for advanced/metastatic disease with low PD-L1 levels TPS-49 % were administered a single dose of sasanlimab 225 mg Q3W subcutaneously along with BID oral dose of 5 mg axitinib on Day 1 of each cycle and Q3W IV infusion of 1 mg/kg SEA-TGT on Day 1 of each cycle during each 21-day cycle.
- Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg): Participants with NSCLC with who were treatment-naïve for advanced/metastatic disease with high PD-L1 (TPS >=50%) were administered a single dose of sasanlimab 225 mg Q3W subcutaneously along with BID oral dose of 5 mg axitinib on Day 1 of each cycle and Q3W IV infusion of 1 mg/kg SEA+ TGT on Day 1 of each cycle during each 21-day cycle.
- Total: Total of all reporting groups
Arm/Group | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg) | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg) | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Total
Number analyzed (Participants) | 4 | 9 | 3 | 6 | 3 | 2 | 7 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 5 | 0 | 1 | 1 | 0 | 5 | 13
  >=65 years | 3 | 4 | 3 | 5 | 2 | 2 | 2 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 1 | 1 | 1 | 2 | 12
  Male | 1 | 6 | 2 | 5 | 2 | 1 | 5 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 4 | 8 | 3 | 6 | 3 | 2 | 6 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 5 | 0 | 1 | 0 | 0 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 4
  White | 2 | 4 | 3 | 3 | 2 | 2 | 7 | 23
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b of Sub-Study A: Percentage of Participants With Dose-Limiting Toxicities (DLT)
Description: DLT=AEs in DLT observation period (OP) related to any study intervention:Grade (G)4 neutropenia;thrombocytopenia or anemia;febrile neutropenia;neutropenic infection;G3 thrombocytopenia with bleeding. Any G>=3 toxicity (except transient G3 fatigue, local reactions/headache that resolved to G<=1/baseline; G3 nausea, vomiting controlled within 72 hrs, G3 hypertension controlled by medical therapy (MT), G3 diarrhea that improved to G<=2 within 72 hrs, G3 skin toxicity that resolved to G<=1 in <7 days after MT, G3 endocrinopathies controlled by MT and tumors flare); Non-hematologic G3 lab abnormality [LA](medical intervention or hospitalization), or any G4 LA;ALT/AST>3*ULN (normal at baseline) or >3*ULN and doubling baseline (>ULN at baseline) and associated with total bilirubin(TB) >2*ULN;or ALT/AST>5*ULN; or TB>3*ULN. Missing 75% of planned doses during DLT OP due to treatment-related toxicities. AE not listed/DLT criteria outside DLT OP was DLT at discretion of sponsor and investigator.
Time Frame: Day 1 up to Day 28 of Cycle 1
Population: DLT-evaluable analysis set included all participants who received at least 1 dose of study treatment in Phase 1b and either experienced DLT during the DLT-observation period or completed the DLT-observation period without DLT.
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg)
Number analyzed (Participants) | 4 | 9
Percentage of participants | 0 | 33.3

2. Primary Outcome: Phase 2 of Sub-Study A: Durable Objective Response Rate (ORR)
Description: Durable ORR was defined as percentage of participants with confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 based on investigator assessment, lasting for at least 10 months from the date of first CR or PR until the date of the first documentation of disease progression (PD), death, or start of new anticancer therapy. CR was defined as complete disappearance of all target lesions with exception of nodal disease. All target nodes must decrease to normal size (short axis <10 millimeter [mm]). PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. PD was defined as 20% increase in sum of diameters of target measurable lesions above smallest sum observed (over baseline if no decrease in the sum was observed during therapy), with a minimum absolute increase of 5 mm.
Time Frame: From the date of first CR or PR until the date of the first documentation of PD, death, or start of new anticancer therapy
Population: Due to a business decision, no participant was enrolled in Phase 2 of sub-study A. Hence, Phase 2 was not initiated and no data was collected.
Groups:
- Phase 2: Sasanlimab + Encorafenib + Binimetinib: Participants with NSCLC with BRAFV600 mutations were planned to receive a combination of sasanlimab encorafenib and binimetinib at the recommended Phase 2 dose.
Arm/Group | Phase 2: Sasanlimab + Encorafenib + Binimetinib
Number analyzed (Participants) | 0

3. Primary Outcome: Phase 1b of Sub-Study B: Percentage of Participants With DLT
Description: DLT=AEs in DLT OP related to any study intervention: G4 neutropenia; thrombocytopenia or anemia; neutropenia; neutropenic infection; G3 thrombocytopenia with bleeding. Any G>=3 toxicity (except transient G3 fatigue, local reactions/headache that resolved to G<=1/baseline; G3 nausea, vomiting controlled within 72 hrs, G3 hypertension controlled by MT, G3 diarrhea that improved to G<=2 within 72 hrs, G3 skin toxicity that resolved to G<=1 in <7 days after MT, G3 endocrinopathies controlled by MT and tumors flare); Non-hematologic G3 LA (medical intervention or hospitalization), or any G4 LA;ALT/AST>3*ULN (normal at baseline) or >3*ULN and doubling baseline (>ULN at baseline) and associated with TB >2*ULN; or ALT/AST>5*ULN; or TB>3*ULN. Missing 75% of planned doses during DLT OP due to treatment-related toxicities. AE not listed/DLT criteria outside DLT OP was DLT at discretion of sponsor and investigator.
Time Frame: Day 1 up to Day 21 of Cycle 1
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg)
Number analyzed (Participants) | 3 | 6
Percentage of participants | 0 | 1

4. Primary Outcome: Phase 2 Sub-Study B: Objective Response Rate
Description: ORR was defined as percentage of participants with confirmed CR or PR according to RECIST v1.1 based on investigator assessment, from the date of first CR or PR until the date of the first documentation of PD, death, or start of new anticancer therapy. CR was defined as complete disappearance of all target lesions with exception of nodal disease. All target nodes must decrease to normal size (short axis <10 millimeter [mm]). PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. PD was defined as 20% increase in sum of diameters of target measurable lesions above smallest sum observed (over baseline if no decrease in the sum was observed during therapy), with a minimum absolute increase of 5 mm.
Time Frame: From the date of first CR or PR until the date of the first documentation of PD, death, or start of new anticancer therapy (maximum of 21 months)
Population: Full analysis set included all participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
Number analyzed (Participants) | 3 | 2 | 7
Percentage of participants | 33.3 [0.8 to 90.6] | 0 [0.0 to 84.2] | 14.3 [0.4 to 57.9]

5. Secondary Outcome: Phase 1b of Sub-Study A: Number of Participants With Adverse Events (AEs) Graded According to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. AEs was graded by the investigator according to NCI CTCAE grade 1 to 5 version 5.0; where Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life-threatening and Grade 5=death.
Time Frame: From the start of study treatment (Cycle1 Day1) up to 30 days after last dose of study treatment (maximum exposure = 38.66 months; maximum follow-up approximately 39.66 months)
Population: Safety analysis set includes all participants who receive at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg)
Number analyzed (Participants) | 4 | 9
Participants
  Grade 1 | 1 | 0
  Grade 2 | 0 | 2
  Grade 3 | 3 | 4
  Grade 4 | 0 | 2
  Grade 5 | 0 | 1

6. Secondary Outcome: Phase 2 of Sub-Study A: Number of Participants With Adverse Events Graded According to NCI-CTCAE Version 5.0
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. AEs were planned to be graded by the investigator according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version (v) 5.0; where Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life-threatening and Grade 5=death.
Time Frame: From the start of study treatment (Cycle1 Day1) up to 30 days after last dose of study treatment
Population: as for outcome 2
Arm/Group | Phase 2: Sasanlimab + Encorafenib + Binimetinib
Number analyzed (Participants) | 0

7. Secondary Outcome: Phase 1b of Sub-Study A: Number of Participants With Shift From Baseline in Hematology Parameters Values Based on CTCAE V5.0
Description: Hematology parameters included: anemia, hemoglobin increased, leukocytosis, lymphocyte count decreased, lymphocyte count increased, leukocytosis, neutrophil count decreased, platelet count decreased, white blood cell decreased. Laboratory abnormalities were graded as per NCI- CTCAE v 5.0 where, grade(G) 0= non-missing lab value that does not meet either of G1 through 4 criteria, G1=mild, G2=moderate, G3=severe and G4= life-threatening or disabling. Baseline is defined as the last assessment prior to the date/time of the first dose of study treatment. Number of participants with shift from baseline in hematology parameters by grades (as per CTCAE version 5.0) were reported.
Time Frame: as for outcome 5
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg)
Number analyzed (Participants) | 4 | 9
Participants
  Anemia: Grade 0 to 0 | 3 | 2
  Anemia: Grade 0 to 1 | 0 | 2
  Anemia: Grade 0 to 2 | 0 | 1
  Anemia: Grade 0 to 3 | 0 | 0
  Anemia: Grade 0 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is not applicable (NA) for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 1 to 0 | 0 | 0
  Anemia: Grade 1 to 1 | 0 | 4
  Anemia: Grade 1 to 2 | 1 | 0
  Anemia: Grade 1 to 3 | 0 | 0
  Anemia: Grade 1 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 2 to 0 | 0 | 0
  Anemia: Grade 2 to 1 | 0 | 0
  Anemia: Grade 2 to 2 | 0 | 0
  Anemia: Grade 2 to 3 | 0 | 0
  Anemia: Grade 2 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 3 to 0 | 0 | 0
  Anemia: Grade 3 to 1 | 0 | 0
  Anemia: Grade 3 to 2 | 0 | 0
  Anemia: Grade 3 to 3 | 0 | 0
  Anemia: Grade 3 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 4 to 0 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 4 to 1 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 4 to 2 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 4 to 3 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 4 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Hemoglobin increased: Grade 0 to 0 | 4 | 8
  Hemoglobin increased: Grade 0 to 1 | 0 | 1
  Hemoglobin increased: Grade 0 to 2 | 0 | 0
  Hemoglobin increased: Grade 0 to 3 | 0 | 0
  Hemoglobin increased: Grade 0 to 4 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 1 to 0 | 0 | 0
  Hemoglobin increased: Grade 1 to 1 | 0 | 0
  Hemoglobin increased: Grade 1 to 2 | 0 | 0
  Hemoglobin increased: Grade 1 to 3 | 0 | 0
  Hemoglobin increased: Grade 1 to 4 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 2 to 0 | 0 | 0
  Hemoglobin increased: Grade 2 to 1 | 0 | 0
  Hemoglobin increased: Grade 2 to 2 | 0 | 0
  Hemoglobin increased: Grade 2 to 3 | 0 | 0
  Hemoglobin increased: Grade 2 to 4 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 3 to 0 | 0 | 0
  Hemoglobin increased: Grade 3 to 1 | 0 | 0
  Hemoglobin increased: Grade 3 to 2 | 0 | 0
  Hemoglobin increased: Grade 3 to 3 | 0 | 0
  Hemoglobin increased: Grade 3 to 4 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 4 to 0 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 4 to 1 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 4 to 2 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 4 to 3 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 4 to 4 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Leukocytosis: Grade 0 to 0 | 4 | 9
  Leukocytosis: Grade 0 to 1 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 0 to 2 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 0 to 3 | 0 | 0
  Leukocytosis: Grade 0 to 4 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 1 to 0 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 1 to 1 | NA — Grade 1 and Gade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 1 to 2 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 1 to 3 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 1 to 4 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 2 to 0 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 2 to 1 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 2 to 2 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 2 to 3 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 2 to 4 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 3 to 0 | 0 | 0
  Leukocytosis: Grade 3 to 1 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 3 to 2 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 3 to 3 | 0 | 0
  Leukocytosis: Grade 3 to 4 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 4 to 0 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 4 to 1 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 4 to 2 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 4 to 3 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 4 to 4 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Lymphocyte count decreased: Grade 0 to 0 | 2 | 3
  Lymphocyte count decreased: Grade 0 to 1 | 1 | 1
  Lymphocyte count decreased: Grade 0 to 2 | 1 | 2
  Lymphocyte count decreased: Grade 0 to 3 | 0 | 0
  Lymphocyte count decreased: Grade 0 to 4 | 0 | 1
  Lymphocyte count decreased: Grade 1 to 0 | 0 | 0
  Lymphocyte count decreased: Grade 1 to 1 | 0 | 0
  Lymphocyte count decreased: Grade 1 to 2 | 0 | 1
  Lymphocyte count decreased: Grade 1 to 3 | 0 | 0
  Lymphocyte count decreased: Grade 1 to 4 | 0 | 0
  Lymphocyte count decreased: Grade 2 to 0 | 0 | 0
  Lymphocyte count decreased: Grade 2 to 1 | 0 | 0
  Lymphocyte count decreased: Grade 2 to 2 | 0 | 1
  Lymphocyte count decreased: Grade 2 to 3 | 0 | 0
  Lymphocyte count decreased: Grade 2 to 4 | 0 | 0
  Lymphocyte count decreased: Grade 3 to 0 | 0 | 0
  Lymphocyte count decreased: Grade 3 to 1 | 0 | 0
  Lymphocyte count decreased: Grade 3 to 2 | 0 | 0
  Lymphocyte count decreased: Grade 3 to 3 | 0 | 0
  Lymphocyte count decreased: Grade 3 to 4 | 0 | 0
  Lymphocyte count decreased: Grade 4 to 0 | 0 | 0
  Lymphocyte count decreased: Grade 4 to 1 | 0 | 0
  Lymphocyte count decreased: Grade 4 to 2 | 0 | 0
  Lymphocyte count decreased: Grade 4 to 3 | 0 | 0
  Lymphocyte count decreased: Grade 4 to 4 | 0 | 0
  Lymphocyte count increased: Grade 0 to 0 | 4 | 9
  Lymphocyte count increased: Grade 0 to 1 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 0 to 2 | 0 | 0
  Lymphocyte count increased: Grade 0 to 3 | 0 | 0
  Lymphocyte count increased: Grade 0 to 4 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 1 to 0 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 1 to 1 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 1 to 2 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 1 to 3 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 1 to 4 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 2 to 0 | 0 | 0
  Lymphocyte count increased: Grade 2 to 1 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 2 to 2 | 0 | 0
  Lymphocyte count increased: Grade 2 to 3 | 0 | 0
  Lymphocyte count increased: Grade 2 to 4 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 3 to 0 | 0 | 0
  Lymphocyte count increased: Grade 3 to 1 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 3 to 2 | 0 | 0
  Lymphocyte count increased: Grade 3 to 3 | 0 | 0
  Lymphocyte count increased: Grade 3 to 4 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 4 to 0 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 4 to 1 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 4 to 2 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 4 to 3 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 4 to 4 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Neutrophil count decreased: Grade 0 to 0 | 4 | 7
  Neutrophil count decreased: Grade 0 to 1 | 0 | 1
  Neutrophil count decreased: Grade 0 to 2 | 0 | 1
  Neutrophil count decreased: Grade 0 to 3 | 0 | 0
  Neutrophil count decreased: Grade 0 to 4 | 0 | 0
  Neutrophil count decreased: Grade 1 to 0 | 0 | 0
  Neutrophil count decreased: Grade 1 to 1 | 0 | 0
  Neutrophil count decreased: Grade 1 to 2 | 0 | 0
  Neutrophil count decreased: Grade 1 to 3 | 0 | 0
  Neutrophil count decreased: Grade 1 to 4 | 0 | 0
  Neutrophil count decreased: Grade 2 to 0 | 0 | 0
  Neutrophil count decreased: Grade 2 to 1 | 0 | 0
  Neutrophil count decreased: Grade 2 to 2 | 0 | 0
  Neutrophil count decreased: Grade 2 to 3 | 0 | 0
  Neutrophil count decreased: Grade 2 to 4 | 0 | 0
  Neutrophil count decreased: Grade 3 to 0 | 0 | 0
  Neutrophil count decreased: Grade 3 to 1 | 0 | 0
  Neutrophil count decreased: Grade 3 to 2 | 0 | 0
  Neutrophil count decreased: Grade 3 to 3 | 0 | 0
  Neutrophil count decreased: Grade 3 to 4 | 0 | 0
  Neutrophil count decreased: Grade 4 to 0 | 0 | 0
  Neutrophil count decreased: Grade 4 to 1 | 0 | 0
  Neutrophil count decreased: Grade 4 to 2 | 0 | 0
  Neutrophil count decreased: Grade 4 to 3 | 0 | 0
  Neutrophil count decreased: Grade 4 to 4 | 0 | 0
  Platelet count decreased: Grade 0 to 0 | 4 | 7
  Platelet count decreased: Grade 0 to 1 | 0 | 1
  Platelet count decreased: Grade 0 to 2 | 0 | 0
  Platelet count decreased: Grade 0 to 3 | 0 | 0
  Platelet count decreased: Grade 0 to 4 | 0 | 0
  Platelet count decreased: Grade 1 to 0 | 0 | 0
  Platelet count decreased: Grade 1 to 1 | 0 | 0
  Platelet count decreased: Grade 1 to 2 | 0 | 1
  Platelet count decreased: Grade 1 to 3 | 0 | 0
  Platelet count decreased: Grade 1 to 4 | 0 | 0
  Platelet count decreased: Grade 2 to 0 | 0 | 0
  Platelet count decreased: Grade 2 to 1 | 0 | 0
  Platelet count decreased: Grade 2 to 2 | 0 | 0
  Platelet count decreased: Grade 2 to 3 | 0 | 0
  Platelet count decreased: Grade 2 to 4 | 0 | 0
  Platelet count decreased: Grade 3 to 0 | 0 | 0
  Platelet count decreased: Grade 3 to 1 | 0 | 0
  Platelet count decreased: Grade 3 to 2 | 0 | 0
  Platelet count decreased: Grade 3 to 3 | 0 | 0
  Platelet count decreased: Grade 3 to 4 | 0 | 0
  Platelet count decreased: Grade 4 to 0 | 0 | 0
  Platelet count decreased: Grade 4 to 1 | 0 | 0
  Platelet count decreased: Grade 4 to 2 | 0 | 0
  Platelet count decreased: Grade 4 to 3 | 0 | 0
  Platelet count decreased: Grade 4 to 4 | 0 | 0
  White blood cell decreased: Grade 0 to 0 | 3 | 8
  White blood cell decreased: Grade 0 to 1 | 1 | 0
  White blood cell decreased: Grade 0 to 2 | 0 | 0
  White blood cell decreased: Grade 0 to 3 | 0 | 0
  White blood cell decreased: Grade 0 to 4 | 0 | 0
  White blood cell decreased: Grade 1 to 0 | 0 | 0
  White blood cell decreased: Grade 1 to 1 | 0 | 0
  White blood cell decreased: Grade 1 to 2 | 0 | 0
  White blood cell decreased: Grade 1 to 3 | 0 | 00
  White blood cell decreased: Grade 1 to 4 | 0 | 0
  White blood cell decreased: Grade 2 to 0 | 0 | 0
  White blood cell decreased: Grade 2 to 1 | 0 | 0
  White blood cell decreased: Grade 2 to 2 | 0 | 1
  White blood cell decreased: Grade 2 to 3 | 0 | 0
  White blood cell decreased: Grade 2 to 4 | 0 | 0
  White blood cell decreased: Grade 3 to 0 | 0 | 0
  White blood cell decreased: Grade 3 to 1 | 0 | 0
  White blood cell decreased: Grade 3 to 2 | 0 | 0
  White blood cell decreased: Grade 3 to 3 | 0 | 0
  White blood cell decreased: Grade 3 to 4 | 0 | 0
  White blood cell decreased: Grade 4 to 0 | 0 | 0
  White blood cell decreased: Grade 4 to 1 | 0 | 0
  White blood cell decreased: Grade 4 to 2 | 0 | 0
  White blood cell decreased: Grade 4 to 3 | 0 | 0
  White blood cell decreased: Grade 4 to 4 | 0 | 0

8. Secondary Outcome: Phase 1b of Sub-Study A: Number of Participants With Shift From Baseline in Chemistry Parameters Values Based on CTCAE V5.0
Description: Chemistry parameters included: alanine aminotransferase (ALT) increase, alkaline phosphatase (ALP) increased, aspartate aminotransferase (AST) increased, blood bilirubin increased, creatinine phosphokinase (CPK) increased, chronic kidney disease (CKD), creatinine increased, hypercalcemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, hyponatremia, lipase increased, serum amylase increased. Chemistry abnormalities were graded as per NCI- CTCAE v 5.0 where, grade(G) 0= non-missing lab value that does not meet either of G1 through 4 criteria, G1=mild, G2=moderate, G3=severe and G4= life-threatening or disabling. Baseline is defined as the last assessment prior to the date/time of the first dose of study treatment. Number of participants with shift from baseline in hematology parameters by grades (as per CTCAE version 5.0) were reported.
Time Frame: as for outcome 5
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg)
Number analyzed (Participants) | 4 | 9
Participants
  Alanine aminotransferase increased: Grade 0 to 0 | 2 | 2
  Alanine aminotransferase increased: Grade 0 to 1 | 2 | 2
  Alanine aminotransferase increased: Grade 0 to 2 | 0 | 2
  Alanine aminotransferase increased: Grade 0 to 3 | 0 | 3
  Alanine aminotransferase increased: Grade 0 to 4 | 0 | 0
  Alanine aminotransferase increased: Grade 1 to 0 | 0 | 0
  Alanine aminotransferase increased: Grade 1 to 1 | 0 | 0
  Alanine aminotransferase increased: Grade 1 to 2 | 0 | 0
  Alanine aminotransferase increased: Grade 1 to 3 | 0 | 0
  Alanine aminotransferase increased: Grade 1 to 4 | 0 | 0
  Alanine aminotransferase increased: Grade 2 to 0 | 0 | 0
  Alanine aminotransferase increased: Grade 2 to 1 | 0 | 0
  Alanine aminotransferase increased: Grade 2 to 2 | 0 | 0
  Alanine aminotransferase increased: Grade 2 to 3 | 0 | 0
  Alanine aminotransferase increased: Grade 2 to 4 | 0 | 0
  Alanine aminotransferase increased: Grade 3 to 0 | 0 | 0
  Alanine aminotransferase increased: Grade 3 to 1 | 0 | 0
  Alanine aminotransferase increased: Grade 3 to 2 | 0 | 0
  Alanine aminotransferase increased: Grade 3 to 3 | 0 | 0
  Alanine aminotransferase increased: Grade 3 to 4 | 0 | 0
  Alanine aminotransferase increased: Grade 4 to 0 | 0 | 0
  Alanine aminotransferase increased: Grade 4 to 1 | 0 | 0
  Alanine aminotransferase increased: Grade 4 to 2 | 0 | 0
  Alanine aminotransferase increased: Grade 4 to 3 | 0 | 0
  Alanine aminotransferase increased: Grade 4 to 4 | 0 | 0
  Alkaline phosphatase increased: Grade 0 to 0 | 1 | 3
  Alkaline phosphatase increased: Grade 0 to 1 | 0 | 2
  Alkaline phosphatase increased: Grade 0 to 2 | 0 | 1
  Alkaline phosphatase increased: Grade 0 to 3 | 0 | 0
  Alkaline phosphatase increased: Grade 0 to 4 | 0 | 0
  Alkaline phosphatase increased: Grade 1 to 0 | 2 | 2
  Alkaline phosphatase increased: Grade 1 to 1 | 0 | 0
  Alkaline phosphatase increased: Grade 1 to 2 | 1 | 0
  Alkaline phosphatase increased: Grade 1 to 3 | 0 | 0
  Alkaline phosphatase increased: Grade 1 to 4 | 0 | 0
  Alkaline phosphatase increased: Grade 2 to 0 | 0 | 0
  Alkaline phosphatase increased: Grade 2 to 1 | 0 | 0
  Alkaline phosphatase increased: Grade 2 to 2 | 0 | 0
  Alkaline phosphatase increased: Grade 2 to 3 | 0 | 0
  Alkaline phosphatase increased: Grade 2 to 4 | 0 | 0
  Alkaline phosphatase increased: Grade 3 to 0 | 0 | 1
  Alkaline phosphatase increased: Grade 3 to 1 | 0 | 0
  Alkaline phosphatase increased: Grade 3 to 2 | 0 | 0
  Alkaline phosphatase increased: Grade 3 to 3 | 0 | 0
  Alkaline phosphatase increased: Grade 3 to 4 | 0 | 0
  Alkaline phosphatase increased: Grade 4 to 0 | 0 | 0
  Alkaline phosphatase increased: Grade 4 to 1 | 0 | 0
  Alkaline phosphatase increased: Grade 4 to 2 | 0 | 0
  Alkaline phosphatase increased: Grade 4 to 3 | 0 | 0
  Alkaline phosphatase increased: Grade 4 to 4 | 0 | 0
  Aspartate aminotransferase increased: Grade 0 to 0 | 2 | 2
  Aspartate aminotransferase increased: Grade 0 to 1 | 2 | 4
  Aspartate aminotransferase increased: Grade 0 to 2 | 0 | 1
  Aspartate aminotransferase increased: Grade 0 to 3 | 0 | 1
  Aspartate aminotransferase increased: Grade 0 to 4 | 0 | 0
  Aspartate aminotransferase increased: Grade 1 to 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 1 to 1 | 0 | 0
  Aspartate aminotransferase increased: Grade 1 to 2 | 0 | 1
  Aspartate aminotransferase increased: Grade 1 to 3 | 0 | 0
  Aspartate aminotransferase increased: Grade 1 to 4 | 0 | 0
  Aspartate aminotransferase increased: Grade 2 to 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 2 to 1 | 0 | 0
  Aspartate aminotransferase increased: Grade 2 to 2 | 0 | 0
  Aspartate aminotransferase increased: Grade 2 to 3 | 0 | 0
  Aspartate aminotransferase increased: Grade 2 to 4 | 0 | 0
  Aspartate aminotransferase increased: Grade 3 to 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 3 to 1 | 0 | 0
  Aspartate aminotransferase increased: Grade 3 to 2 | 0 | 0
  Aspartate aminotransferase increased: Grade 3 to 3 | 0 | 0
  Aspartate aminotransferase increased: Grade 3 to 4 | 0 | 0
  Aspartate aminotransferase increased: Grade 4 to 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 4 to 1 | 0 | 0
  Aspartate aminotransferase increased: Grade 4 to 2 | 0 | 0
  Aspartate aminotransferase increased: Grade 4 to 3 | 0 | 0
  Aspartate aminotransferase increased: Grade 4 to 4 | 0 | 0
  Blood bilirubin increased: Grade 0 to 0 | 4 | 8
  Blood bilirubin increased: Grade 0 to 1 | 0 | 0
  Blood bilirubin increased: Grade 0 to 2 | 0 | 0
  Blood bilirubin increased: Grade 0 to 3 | 0 | 1
  Blood bilirubin increased: Grade 0 to 4 | 0 | 0
  Blood bilirubin increased: Grade 1 to 0 | 0 | 0
  Blood bilirubin increased: Grade 1 to 1 | 0 | 0
  Blood bilirubin increased: Grade 1 to 2 | 0 | 0
  Blood bilirubin increased: Grade 1 to 3 | 0 | 0
  Blood bilirubin increased: Grade 1 to 4 | 0 | 0
  Blood bilirubin increased: Grade 2 to 0 | 0 | 0
  Blood bilirubin increased: Grade 2 to 1 | 0 | 0
  Blood bilirubin increased: Grade 2 to 2 | 0 | 0
  Blood bilirubin increased: Grade 2 to 3 | 0 | 0
  Blood bilirubin increased: Grade 2 to 4 | 0 | 0
  Blood bilirubin increased: Grade 3 to 0 | 0 | 0
  Blood bilirubin increased: Grade 3 to 1 | 0 | 0
  Blood bilirubin increased: Grade 3 to 2 | 0 | 0
  Blood bilirubin increased: Grade 3 to 3 | 0 | 0
  Blood bilirubin increased: Grade 3 to 4 | 0 | 0
  Blood bilirubin increased: Grade 4 to 0 | 0 | 0
  Blood bilirubin increased: Grade 4 to 1 | 0 | 0
  Blood bilirubin increased: Grade 4 to 2 | 0 | 0
  Blood bilirubin increased: Grade 4 to 3 | 0 | 0
  Blood bilirubin increased: Grade 4 to 4 | 0 | 0
  CPK increased: Grade 0 to 0 | 2 | 4
  CPK increased: Grade 0 to 1 | 2 | 1
  CPK increased: Grade 0 to 2 | 0 | 2
  CPK increased: Grade 0 to 3 | 0 | 1
  CPK increased: Grade 0 to 4 | 0 | 1
  CPK increased: Grade 1 to 0 | 0 | 0
  CPK increased: Grade 1 to 1 | 0 | 0
  CPK increased: Grade 1 to 2 | 0 | 0
  CPK increased: Grade 1 to 3 | 0 | 0
  CPK increased: Grade 1 to 4 | 0 | 0
  CPK increased: Grade 2 to 0 | 0 | 0
  CPK increased: Grade 2 to 1 | 0 | 0
  CPK increased: Grade 2 to 2 | 0 | 0
  CPK increased: Grade 2 to 3 | 0 | 0
  CPK increased: Grade 2 to 4 | 0 | 0
  CPK increased: Grade 3 to 0 | 0 | 0
  CPK increased: Grade 3 to 1 | 0 | 0
  CPK increased: Grade 3 to 2 | 0 | 0
  CPK increased: Grade 3 to 3 | 0 | 0
  CPK increased: Grade 3 to 4 | 0 | 0
  CPK increased: Grade 4 to 0 | 0 | 0
  CPK increased: Grade 4 to 1 | 0 | 0
  CPK increased: Grade 4 to 2 | 0 | 0
  CPK increased: Grade 4 to 3 | 0 | 0
  CPK increased: Grade 4 to 4 | 0 | 0
  Chronic kidney disease: Grade 0 to 0 | 1 | 3
  Chronic kidney disease: Grade 0 to 1 | 0 | 1
  Chronic kidney disease: Grade 0 to 2 | 2 | 3
  Chronic kidney disease: Grade 0 to 3 | 0 | 0
  Chronic kidney disease: Grade 0 to 4 | 0 | 0
  Chronic kidney disease: Grade 1 to 0 | 0 | 0
  Chronic kidney disease: Grade 1 to 1 | 1 | 1
  Chronic kidney disease: Grade 1 to 2 | 0 | 0
  Chronic kidney disease: Grade 1 to 3 | 0 | 0
  Chronic kidney disease: Grade 1 to 4 | 0 | 0
  Chronic kidney disease: Grade 2 to 0 | 0 | 0
  Chronic kidney disease: Grade 2 to 1 | 0 | 0
  Chronic kidney disease: Grade 2 to 2 | 0 | 1
  Chronic kidney disease: Grade 2 to 3 | 0 | 0
  Chronic kidney disease: Grade 2 to 4 | 0 | 0
  Chronic kidney disease: Grade 3 to 0 | 0 | 0
  Chronic kidney disease: Grade 3 to 1 | 0 | 0
  Chronic kidney disease: Grade 3 to 2 | 0 | 0
  Chronic kidney disease: Grade 3 to 3 | 0 | 0
  Chronic kidney disease: Grade 3 to 4 | 0 | 0
  Chronic kidney disease: Grade 4 to 0 | 0 | 0
  Chronic kidney disease: Grade 4 to 1 | 0 | 0
  Chronic kidney disease: Grade 4 to 2 | 0 | 0
  Chronic kidney disease: Grade 4 to 3 | 0 | 0
  Chronic kidney disease: Grade 4 to 4 | 0 | 0
  Creatinine increased: Grade 0 to 0 | 1 | 6
  Creatinine increased: Grade 0 to 1 | 2 | 2
  Creatinine increased: Grade 0 to 2 | 1 | 1
  Creatinine increased: Grade 0 to 3 | 0 | 0
  Creatinine increased: Grade 0 to 4 | 0 | 0
  Creatinine increased: Grade 1 to 0 | 0 | 0
  Creatinine increased: Grade 1 to 1 | 0 | 0
  Creatinine increased: Grade 1 to 2 | 0 | 0
  Creatinine increased: Grade 1 to 3 | 0 | 0
  Creatinine increased: Grade 1 to 4 | 0 | 0
  Creatinine increased: Grade 2 to 0 | 0 | 0
  Creatinine increased: Grade 2 to 1 | 0 | 0
  Creatinine increased: Grade 2 to 2 | 0 | 0
  Creatinine increased: Grade 2 to 3 | 0 | 0
  Creatinine increased: Grade 2 to 4 | 0 | 0
  Creatinine increased: Grade 3 to 0 | 0 | 0
  Creatinine increased: Grade 3 to 1 | 0 | 0
  Creatinine increased: Grade 3 to 2 | 0 | 0
  Creatinine increased: Grade 3 to 3 | 0 | 0
  Creatinine increased: Grade 3 to 4 | 0 | 0
  Creatinine increased: Grade 4 to 0 | 0 | 0
  Creatinine increased: Grade 4 to 1 | 0 | 0
  Creatinine increased: Grade 4 to 2 | 0 | 0
  Creatinine increased: Grade 4 to 3 | 0 | 0
  Creatinine increased: Grade 4 to 4 | 0 | 0
  Hypercalcemia: Grade 0 to 0 | 3 | 4
  Hypercalcemia: Grade 0 to 1 | 1 | 5
  Hypercalcemia: Grade 0 to 2 | 0 | 0
  Hypercalcemia: Grade 0 to 3 | 0 | 0
  Hypercalcemia: Grade 0 to 4 | 0 | 0
  Hypercalcemia: Grade 1 to 0 | 0 | 0
  Hypercalcemia: Grade 1 to 1 | 0 | 0
  Hypercalcemia: Grade 1 to 2 | 0 | 0
  Hypercalcemia: Grade 1 to 3 | 0 | 0
  Hypercalcemia: Grade 1 to 4 | 0 | 0
  Hypercalcemia: Grade 2 to 0 | 0 | 0
  Hypercalcemia: Grade 2 to 1 | 0 | 0
  Hypercalcemia: Grade 2 to 2 | 0 | 0
  Hypercalcemia: Grade 2 to 3 | 0 | 0
  Hypercalcemia: Grade 2 to 4 | 0 | 0
  Hypercalcemia: Grade 3 to 0 | 0 | 0
  Hypercalcemia: Grade 3 to 1 | 0 | 0
  Hypercalcemia: Grade 3 to 2 | 0 | 0
  Hypercalcemia: Grade 3 to 3 | 0 | 0
  Hypercalcemia: Grade 3 to 4 | 0 | 0
  Hypercalcemia: Grade 4 to 0 | 0 | 0
  Hypercalcemia: Grade 4 to 1 | 0 | 0
  Hypercalcemia: Grade 4 to 2 | 0 | 0
  Hypercalcemia: Grade 4 to 3 | 0 | 0
  Hypercalcemia: Grade 4 to 4 | 0 | 0
  Hyperkalemia: Grade 0 to 0 | 4 | 8
  Hyperkalemia: Grade 0 to 1 | 0 | 1
  Hyperkalemia: Grade 0 to 2 | 0 | 0
  Hyperkalemia: Grade 0 to 3 | 0 | 0
  Hyperkalemia: Grade 0 to 4 | 0 | 0
  Hyperkalemia: Grade 1 to 0 | 0 | 0
  Hyperkalemia: Grade 1 to 1 | 0 | 0
  Hyperkalemia: Grade 1 to 2 | 0 | 0
  Hyperkalemia: Grade 1 to 3 | 0 | 0
  Hyperkalemia: Grade 1 to 4 | 0 | 0
  Hyperkalemia: Grade 2 to 0 | 0 | 0
  Hyperkalemia: Grade 2 to 1 | 0 | 0
  Hyperkalemia: Grade 2 to 2 | 0 | 0
  Hyperkalemia: Grade 2 to 3 | 0 | 0
  Hyperkalemia: Grade 2 to 4 | 0 | 0
  Hyperkalemia: Grade 3 to 0 | 0 | 0
  Hyperkalemia: Grade 3 to 1 | 0 | 0
  Hyperkalemia: Grade 3 to 2 | 0 | 0
  Hyperkalemia: Grade 3 to 3 | 0 | 0
  Hyperkalemia: Grade 3 to 4 | 0 | 0
  Hyperkalemia: Grade 4 to 0 | 0 | 0
  Hyperkalemia: Grade 4 to 1 | 0 | 0
  Hyperkalemia: Grade 4 to 2 | 0 | 0
  Hyperkalemia: Grade 4 to 3 | 0 | 0
  Hyperkalemia: Grade 4 to 4 | 0 | 0
  Hypermagnesemia: Grade 0 to 0 | 4 | 8
  Hypermagnesemia: Grade 0 to 1 | 0 | 1
  Hypermagnesemia: Grade 0 to 2 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 0 to 3 | 0 | 0
  Hypermagnesemia: Grade 0 to 4 | 0 | 0
  Hypermagnesemia: Grade 1 to 0 | 0 | 0
  Hypermagnesemia: Grade 1 to 1 | 0 | 0
  Hypermagnesemia: Grade 1 to 2 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 1 to 3 | 0 | 0
  Hypermagnesemia: Grade 1 to 4 | 0 | 0
  Hypermagnesemia: Grade 2 to 0 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 2 to 1 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 2 to 2 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 2 to 3 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 2 to 4 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 3 to 0 | 0 | 0
  Hypermagnesemia: Grade 3 to 1 | 0 | 0
  Hypermagnesemia: Grade 3 to 2 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 3 to 3 | 0 | 0
  Hypermagnesemia: Grade 3 to 4 | 0 | 0
  Hypermagnesemia: Grade 4 to 0 | 0 | 0
  Hypermagnesemia: Grade 4 to 1 | 0 | 0
  Hypermagnesemia: Grade 4 to 2 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 4 to 3 | 0 | 0
  Hypermagnesemia: Grade 4 to 4 | 0 | 0
  Hypernatremia: Grade 0 to 0 | 4 | 8
  Hypernatremia: Grade 0 to 1 | 0 | 1
  Hypernatremia: Grade 0 to 2 | 0 | 0
  Hypernatremia: Grade 0 to 3 | 0 | 0
  Hypernatremia: Grade 0 to 4 | 0 | 0
  Hypernatremia: Grade 1 to 0 | 0 | 0
  Hypernatremia: Grade 1 to 1 | 0 | 0
  Hypernatremia: Grade 1 to 2 | 0 | 0
  Hypernatremia: Grade 1 to 3 | 0 | 0
  Hypernatremia: Grade 1 to 4 | 0 | 0
  Hypernatremia: Grade 2 to 0 | 0 | 0
  Hypernatremia: Grade 2 to 1 | 0 | 0
  Hypernatremia: Grade 2 to 2 | 0 | 0
  Hypernatremia: Grade 2 to 3 | 0 | 0
  Hypernatremia: Grade 2 to 4 | 0 | 0
  Hypernatremia: Grade 3 to 0 | 0 | 0
  Hypernatremia: Grade 3 to 1 | 0 | 0
  Hypernatremia: Grade 3 to 2 | 0 | 0
  Hypernatremia: Grade 3 to 3 | 0 | 0
  Hypernatremia: Grade 3 to 4 | 0 | 0
  Hypernatremia: Grade 4 to 0 | 0 | 0
  Hypernatremia: Grade 4 to 1 | 0 | 0
  Hypernatremia: Grade 4 to 2 | 0 | 0
  Hypernatremia: Grade 4 to 3 | 0 | 0
  Hypernatremia: Grade 4 to 4 | 0 | 0
  Hypoalbuminemia: Grade 0 to 0 | 2 | 3
  Hypoalbuminemia: Grade 0 to 1 | 1 | 3
  Hypoalbuminemia: Grade 0 to 2 | 0 | 1
  Hypoalbuminemia: Grade 0 to 3 | 1 | 0
  Hypoalbuminemia: Grade 0 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 1 to 0 | 0 | 0
  Hypoalbuminemia: Grade 1 to 1 | 0 | 1
  Hypoalbuminemia: Grade 1 to 2 | 0 | 1
  Hypoalbuminemia: Grade 1 to 3 | 0 | 0
  Hypoalbuminemia: Grade 1 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 2 to 0 | 0 | 0
  Hypoalbuminemia: Grade 2 to 1 | 0 | 0
  Hypoalbuminemia: Grade 2 to 2 | 0 | 0
  Hypoalbuminemia: Grade 2 to 3 | 0 | 0
  Hypoalbuminemia: Grade 2 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 3 to 0 | 0 | 0
  Hypoalbuminemia: Grade 3 to 1 | 0 | 0
  Hypoalbuminemia: Grade 3 to 2 | 0 | 0
  Hypoalbuminemia: Grade 3 to 3 | 0 | 0
  Hypoalbuminemia: Grade 3 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 4 to 0 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 4 to 1 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 4 to 2 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 4 to 3 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 4 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypocalcemia: Grade 0 to 0 | 4 | 7
  Hypocalcemia: Grade 0 to 1 | 0 | 2
  Hypocalcemia: Grade 0 to 2 | 0 | 0
  Hypocalcemia: Grade 0 to 3 | 0 | 0
  Hypocalcemia: Grade 0 to 4 | 0 | 0
  Hypocalcemia: Grade 1 to 0 | 0 | 0
  Hypocalcemia: Grade 1 to 1 | 0 | 0
  Hypocalcemia: Grade 1 to 2 | 0 | 0
  Hypocalcemia: Grade 1 to 3 | 0 | 0
  Hypocalcemia: Grade 1 to 4 | 0 | 0
  Hypocalcemia: Grade 2 to 0 | 0 | 0
  Hypocalcemia: Grade 2 to 1 | 0 | 0
  Hypocalcemia: Grade 2 to 2 | 0 | 0
  Hypocalcemia: Grade 2 to 3 | 0 | 0
  Hypocalcemia: Grade 2 to 4 | 0 | 0
  Hypocalcemia: Grade 3 to 0 | 0 | 0
  Hypocalcemia: Grade 3 to 1 | 0 | 0
  Hypocalcemia: Grade 3 to 2 | 0 | 0
  Hypocalcemia: Grade 3 to 3 | 0 | 0
  Hypocalcemia: Grade 3 to 4 | 0 | 0
  Hypocalcemia: Grade 4 to 0 | 0 | 0
  Hypocalcemia: Grade 4 to 1 | 0 | 0
  Hypocalcemia: Grade 4 to 2 | 0 | 0
  Hypocalcemia: Grade 4 to 3 | 0 | 0
  Hypocalcemia: Grade 4 to 4 | 0 | 0
  Hypoglycemia: Grade 0 to 0 | 4 | 7
  Hypoglycemia: Grade 0 to 1 | 0 | 1
  Hypoglycemia: Grade 0 to 2 | 0 | 0
  Hypoglycemia: Grade 0 to 3 | 0 | 0
  Hypoglycemia: Grade 0 to 4 | 0 | 0
  Hypoglycemia: Grade 1 to 0 | 0 | 1
  Hypoglycemia: Grade 1 to 1 | 0 | 0
  Hypoglycemia: Grade 1 to 2 | 0 | 0
  Hypoglycemia: Grade 1 to 3 | 0 | 0
  Hypoglycemia: Grade 1 to 4 | 0 | 0
  Hypoglycemia: Grade 2 to 0 | 0 | 0
  Hypoglycemia: Grade 2 to 1 | 0 | 0
  Hypoglycemia: Grade 2 to 2 | 0 | 0
  Hypoglycemia: Grade 2 to 3 | 0 | 0
  Hypoglycemia: Grade 2 to 4 | 0 | 0
  Hypoglycemia: Grade 3 to 0 | 0 | 0
  Hypoglycemia: Grade 3 to 1 | 0 | 0
  Hypoglycemia: Grade 3 to 2 | 0 | 0
  Hypoglycemia: Grade 3 to 3 | 0 | 0
  Hypoglycemia: Grade 3 to 4 | 0 | 0
  Hypoglycemia: Grade 4 to 0 | 0 | 0
  Hypoglycemia: Grade 4 to 1 | 0 | 0
  Hypoglycemia: Grade 4 to 2 | 0 | 0
  Hypoglycemia: Grade 4 to 3 | 0 | 0
  Hypoglycemia: Grade 4 to 4 | 0 | 0
  Hypokalemia: Grade 0 to 0 | 4 | 7
  Hypokalemia: Grade 0 to 1 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 0 to 2 | 0 | 1
  Hypokalemia: Grade 0 to 3 | 0 | 1
  Hypokalemia: Grade 0 to 4 | 0 | 0
  Hypokalemia: Grade 1 to 0 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 1 to 1 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 1 to 2 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 1 to 3 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 1 to 4 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 2 to 0 | 0 | 0
  Hypokalemia: Grade 2 to 1 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 2 to 2 | 0 | 0
  Hypokalemia: Grade 2 to 3 | 0 | 0
  Hypokalemia: Grade 2 to 4 | 0 | 0
  Hypokalemia: Grade 3 to 0 | 0 | 0
  Hypokalemia: Grade 3 to 1 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 3 to 2 | 0 | 0
  Hypokalemia: Grade 3 to 3 | 0 | 0
  Hypokalemia: Grade 3 to 4 | 0 | 0
  Hypokalemia: Grade 4 to 0 | 0 | 0
  Hypokalemia: Grade 4 to 1 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 4 to 2 | 0 | 0
  Hypokalemia: Grade 4 to 3 | 0 | 0
  Hypokalemia: Grade 4 to 4 | 0 | 0
  Hypomagnesemia: Grade 0 to 0 | 4 | 8
  Hypomagnesemia: Grade 0 to 1 | 0 | 1
  Hypomagnesemia: Grade 0 to 2 | 0 | 0
  Hypomagnesemia: Grade 0 to 3 | 0 | 0
  Hypomagnesemia: Grade 0 to 4 | 0 | 0
  Hypomagnesemia: Grade 1 to 0 | 0 | 0
  Hypomagnesemia: Grade 1 to 1 | 0 | 0
  Hypomagnesemia: Grade 1 to 2 | 0 | 0
  Hypomagnesemia: Grade 1 to 3 | 0 | 0
  Hypomagnesemia: Grade 1 to 4 | 0 | 0
  Hypomagnesemia: Grade 2 to 0 | 0 | 0
  Hypomagnesemia: Grade 2 to 1 | 0 | 0
  Hypomagnesemia: Grade 2 to 2 | 0 | 0
  Hypomagnesemia: Grade 2 to 3 | 0 | 0
  Hypomagnesemia: Grade 2 to 4 | 0 | 0
  Hypomagnesemia: Grade 3 to 0 | 0 | 0
  Hypomagnesemia: Grade 3 to 1 | 0 | 0
  Hypomagnesemia: Grade 3 to 2 | 0 | 0
  Hypomagnesemia: Grade 3 to 3 | 0 | 0
  Hypomagnesemia: Grade 3 to 4 | 0 | 0
  Hypomagnesemia: Grade 4 to 0 | 0 | 0
  Hypomagnesemia: Grade 4 to 1 | 0 | 0
  Hypomagnesemia: Grade 4 to 2 | 0 | 0
  Hypomagnesemia: Grade 4 to 3 | 0 | 0
  Hypomagnesemia: Grade 4 to 4 | 0 | 0
  Hyponatremia: Grade 0 to 0 | 3 | 5
  Hyponatremia: Grade 0 to 1 | 0 | 1
  Hyponatremia: Grade 0 to 2 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 0 to 3 | 0 | 1
  Hyponatremia: Grade 0 to 4 | 0 | 0
  Hyponatremia: Grade 1 to 0 | 1 | 0
  Hyponatremia: Grade 1 to 1 | 0 | 0
  Hyponatremia: Grade 1 to 2 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 1 to 3 | 0 | 2
  Hyponatremia: Grade 1 to 4 | 0 | 0
  Hyponatremia: Grade 2 to 0 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 2 to 1 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 2 to 2 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 2 to 3 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 2 to 4 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 3 to 0 | 0 | 0
  Hyponatremia: Grade 3 to 1 | 0 | 0
  Hyponatremia: Grade 3 to 2 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 3 to 3 | 0 | 0
  Hyponatremia: Grade 3 to 4 | 0 | 0
  Hyponatremia: Grade 4 to 0 | 0 | 0
  Hyponatremia: Grade 4 to 1 | 0 | 0
  Hyponatremia: Grade 4 to 2 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 4 to 3 | 0 | 0
  Hyponatremia: Grade 4 to 4 | 0 | 0
  Lipase increased: Grade 0 to 0 | 1 | 5
  Lipase increased: Grade 0 to 1 | 2 | 3
  Lipase increased: Grade 0 to 2 | 1 | 1
  Lipase increased: Grade 0 to 3 | 0 | 0
  Lipase increased: Grade 0 to 4 | 0 | 0
  Lipase increased: Grade 1 to 0 | 0 | 0
  Lipase increased: Grade 1 to 1 | 0 | 0
  Lipase increased: Grade 1 to 2 | 0 | 0
  Lipase increased: Grade 1 to 3 | 0 | 0
  Lipase increased: Grade 1 to 4 | 0 | 0
  Lipase increased: Grade 2 to 0 | 0 | 0
  Lipase increased: Grade 2 to 1 | 0 | 0
  Lipase increased: Grade 2 to 2 | 0 | 0
  Lipase increased: Grade 2 to 3 | 0 | 0
  Lipase increased: Grade 2 to 4 | 0 | 0
  Lipase increased: Grade 3 to 0 | 0 | 0
  Lipase increased: Grade 3 to 1 | 0 | 0
  Lipase increased: Grade 3 to 2 | 0 | 0
  Lipase increased: Grade 3 to 3 | 0 | 0
  Lipase increased: Grade 3 to 4 | 0 | 0
  Lipase increased: Grade 4 to 0 | 0 | 0
  Lipase increased: Grade 4 to 1 | 0 | 0
  Lipase increased: Grade 4 to 2 | 0 | 0
  Lipase increased: Grade 4 to 3 | 0 | 0
  Lipase increased: Grade 4 to 4 | 0 | 0
  Serum amylase increased: Grade 0 to 0 | 4 | 7
  Serum amylase increased: Grade 0 to 1 | 0 | 0
  Serum amylase increased: Grade 0 to 2 | 0 | 0
  Serum amylase increased: Grade 0 to 3 | 0 | 1
  Serum amylase increased: Grade 0 to 4 | 0 | 0
  Serum amylase increased: Grade 1 to 0 | 0 | 0
  Serum amylase increased: Grade 1 to 1 | 0 | 1
  Serum amylase increased: Grade 1 to 2 | 0 | 0
  Serum amylase increased: Grade 1 to 3 | 0 | 0
  Serum amylase increased: Grade 1 to 4 | 0 | 0
  Serum amylase increased: Grade 2 to 0 | 0 | 0
  Serum amylase increased: Grade 2 to 1 | 0 | 0
  Serum amylase increased: Grade 2 to 2 | 0 | 0
  Serum amylase increased: Grade 2 to 3 | 0 | 0
  Serum amylase increased: Grade 2 to 4 | 0 | 0
  Serum amylase increased: Grade 3 to 0 | 0 | 0
  Serum amylase increased: Grade 3 to 1 | 0 | 0
  Serum amylase increased: Grade 3 to 2 | 0 | 0
  Serum amylase increased: Grade 3 to 3 | 0 | 0
  Serum amylase increased: Grade 3 to 4 | 0 | 0
  Serum amylase increased: Grade 4 to 0 | 0 | 0
  Serum amylase increased: Grade 4 to 1 | 0 | 0
  Serum amylase increased: Grade 4 to 2 | 0 | 0
  Serum amylase increased: Grade 4 to 3 | 0 | 0
  Serum amylase increased: Grade 4 to 4 | 0 | 0

9. Secondary Outcome: Phase 2 of Sub-Study A: Number of Participants With Laboratory Abnormalities
Description: Hematology and clinical chemistry parameters were planned to be assessed.
Time Frame: From the start of study treatment (Cycle1 Day1) up to 30 days after last dose of study treatment
Population: as for outcome 2
Arm/Group | Phase 2: Sasanlimab + Encorafenib + Binimetinib
Number analyzed (Participants) | 0

10. Secondary Outcome: Phase 1b of Sub-Study A: Durable Objective Response Rate (ORR)
Description: Durable ORR was defined as percentage of participants with confirmed CR or PR according to RECIST v1.1 based on investigator assessment, lasting for at least 10 months from the date of first CR or PR until the date of the first documentation of PD, death, or start of new anticancer therapy. CR was defined as complete disappearance of all target lesions with exception of nodal disease. All target nodes must decrease to normal size (short axis <10 milli meter [mm]). PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. PD was defined as 20% increase in sum of diameters of target measurable lesions above smallest sum observed (over baseline if no decrease in the sum is observed during therapy) with a minimum absolute increase of 5 mm. Non-CR/Non-PD: Persistence of any non-target lesions and/or tumor marker level (if being followed) above the normal limits.
Time Frame: From the date of first CR or PR until the date of the first documentation of PD, death, or start of new anticancer therapy (approximately 38.66 months)
Population: Full analysis set included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg)
Number analyzed (Participants) | 4 | 9
Percentage of Participants | 25.0 [0.6 to 80.6] | 44.4 [13.7 to 78.8]

11. Secondary Outcome: Phase 1b of Sub-Study A: Objective Response Rate
Description: Objective response rate is defined as percentage of participants with confirmed best overall response of CR or PR according to RECIST v1.1 from the date of first dose of study treatment until the date of the first documentation of PD. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. PD was defined as 20% increase in sum of diameters of target measurable lesions above smallest sum observed (over baseline if no decrease in the sum is observed during therapy) with a minimum absolute increase of 5 mm. Non-CR/Non-PD: Persistence of any non-target lesions and/or tumor marker level (if being followed) above the normal limits.
Time Frame: as for outcome 10
Population: Full analysis set included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg)
Number analyzed (Participants) | 4 | 9
Percentage of Participants | 50.0 [6.8 to 93.2] | 44.4 [13.7 to 78.8]

12. Secondary Outcome: Phase 2 of Sub-Study A: Objective Response Rate
Description: Objective response (OR) rate is defined as percentage of participants with confirmed best overall response of CR or PR according to RECIST v1.1 from the date of first dose of study treatment until the date of the first documentation of PD. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions.
Time Frame: as for outcome 2
Population: as for outcome 2
Arm/Group | Phase 2: Sasanlimab + Encorafenib + Binimetinib
Number analyzed (Participants) | 0

13. Secondary Outcome: Phase 2 of Sub-Study A: Duration of Response (DR)
Description: DR was defined for participants with confirmed OR as time from date of first documentation of OR to the date of first documentation of PD or death (any cause), whichever occurred first. OR=CR or PR according to RECIST v1.1 based on investigator assessment. CR and PR must be confirmed by repeat assessments performed no <4 weeks after criteria for response were first met. CR=complete disappearance of all target lesions (TLs) with exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). PR=greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions (TMLs). PD=20% increase in sum of diameters of TMLs above smallest sum observed (over baseline if no decrease in sum was observed during therapy), with a minimum absolute increase of 5 mm.
Time Frame: From the date of first documentation of OR to the date of the first documentation of PD or death due to any cause, whichever occurred first
Population: as for outcome 2
Arm/Group | Phase 2: Sasanlimab + Encorafenib + Binimetinib
Number analyzed (Participants) | 0

14. Secondary Outcome: Phase 2 of Sub-Study A: Time to Tumor Response (TTR)
Description: TTR is defined for participants with confirmed objective response as the time from the date of first dose of study treatment to the date of first documentation of objective response (CR or PR) which was subsequently confirmed. CR=complete disappearance of all target lesions with exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). PR=greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions.
Time Frame: From the date of first dose of study treatment to the date of first documentation of objective response
Population: as for outcome 2
Groups:
- Phase 2: Sasanlimab + Encorafenib + Binimetinib: Participants with NSCLC with BRAFV600 mutations were planned to receive a combination of sasanlimab, encorafenib and binimetinib at the recommended Phase 2 dose.
Arm/Group | Phase 2: Sasanlimab + Encorafenib + Binimetinib
Number analyzed (Participants) | 0

15. Secondary Outcome: Phase 2 of Sub-Study A: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the date of first dose of study treatment to the date of first documentation of PD or death due to any cause, whichever occurred first. PD=20% increase in sum of diameters of target measurable lesions above smallest sum observed (over baseline if no decrease in sum was observed during therapy), with a minimum absolute increase of 5 mm.
Time Frame: From the date of first dose of study treatment to the date of first documentation of PD or death due to any cause, whichever occurred first
Population: as for outcome 2
Arm/Group | Phase 2: Sasanlimab + Encorafenib + Binimetinib
Number analyzed (Participants) | 0

16. Secondary Outcome: Phase 2 of Sub-Study A: Overall Survival (OS)
Description: OS is defined as the time from the date of first dose of study treatment to the date of death due to any cause. Participants last known to be alive were planned to be censored at the date of last contact.
Time Frame: From the date of first dose of study treatment to the date of death due to any cause or censoring date
Population: as for outcome 2
Arm/Group | Phase 2: Sasanlimab + Encorafenib + Binimetinib
Number analyzed (Participants) | 0

17. Secondary Outcome: Phase 1b of Sub-Study A: Area Under the Concentration Versus Time Curve Over the Dosing Interval (AUCtau) After Single Dose of Sasanlimab
Description: AUCtau was defined as area under the plasma concentration time curve from time zero to the next dose.
Time Frame: Cycle 1 (pre-dose on Day 1, 168 hours [Day 8] and 336 hours [Day 15] and Day 28 post-dose) (1 cycle= 28 days)
Population: Pharmacokinetic (PK) parameter analysis set was subset of safety analysis set (participants who received at least 1 dose of study drug) with participants who had at least 1 of PK parameters of interest for measured analytes related to study drug (i.e., sasanlimab). Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms*hour per milliliter
Arm/Group | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg)
Number analyzed (Participants) | 3 | 7
Micrograms*hour per milliliter | 12500 (65) | 24850 (17)

18. Secondary Outcome: Phase 2 of Sub-Study A: Area Under the Concentration Versus Time Curve Over the Dosing Interval (AUCtau) After Single Dose of Sasanlimab
Time Frame: Cycle 1 (pre-dose on Day 1, 336 hours [Day 15] and Day 28 post-dose) (1 cycle= 28 days)
Population: as for outcome 2
Arm/Group | Phase 2: Sasanlimab + Encorafenib + Binimetinib
Number analyzed (Participants) | 0

19. Secondary Outcome: Phase 1b of Sub-Study A: Maximum Observed Plasma Concentration (Cmax) of Sasanlimab
Time Frame: Cycle 1 (pre-dose on Day 1, 168 hours [Day 8],336 hours [Day 15] and Day 28 post-dose) and Cycle 5 (pre-dose on Day 1 and 168 hours [Day 8] post dose) (1 cycle= 28 days)
Population: PK parameter analysis set was subset of safety analysis set (participants who received at least 1 dose of study drug) with participants who had at least 1 of PK parameters of interest for measured analytes related to study drug (i.e., sasanlimab). Here, 'Number Analyzed' signifies participants evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg)
Number analyzed (Participants) | 4 | 9
Micrograms per milliliter
  Cycle 1 | 29.49 (55) | 45.04 (38)
  Cycle 5: number analyzed (Participants) | 1 | 1
  Cycle 5 | 64.60 (NA) — Geometric Coefficient of Variation could not be calculated as a single participant was analyzed. | 70.90 (NA) — Geometric Coefficient of Variation could not be calculated as a single participant was analyzed.

20. Secondary Outcome: Phase 2 of Sub-Study A: Maximum Observed Plasma Concentration (Cmax) of Sasanlimab
Time Frame: Cycle 1 (pre-dose on Day 1, 336 hours [Day 15] and Day 28 post-dose) and Cycle 5 Day 1 (pre-dose) (1 cycle= 28 days)
Population: as for outcome 2
Arm/Group | Phase 2: Sasanlimab + Encorafenib + Binimetinib
Number analyzed (Participants) | 0

21. Secondary Outcome: Phase 1b of Sub-Study A: Time for Cmax (Tmax) of Sasanlimab
Time Frame: Cycle 1 (pre-dose on Day 1, 168 hours [Day 8], 336 hours [Day 15] and Day 28 post-dose) and Cycle 5 (pre-dose on Day 1 and 168 hours [Day 8] post dose) (1 cycle= 28 days)
Population: as for outcome 19
Measure: Median (Full Range); unit: Hour
Arm/Group | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg)
Number analyzed (Participants) | 4 | 9
Hour
  Cycle 1 | 164 [144 to 168] | 209 [143 to 359]
  Cycle 5: number analyzed (Participants) | 1 | 1
  Cycle 5 | 168 [168 to 168] | 162 [162 to 162]

22. Secondary Outcome: Phase 2 of Sub-Study A: Time for Cmax (Tmax) of Sasanlimab
Time Frame: Cycle 1 (pre-dose on Day 1, 336 hours [Day 15] and Day 28 post-dose) and Cycle 5 Day 1 (pre-dose) (1 cycle= 28 days)
Population: as for outcome 2
Arm/Group | Phase 2: Sasanlimab + Encorafenib + Binimetinib
Number analyzed (Participants) | 0

23. Secondary Outcome: Phase 1b of Sub-Study A: Pre-dose Concentration During Multiple Dosing (Ctrough) of Sasanlimab
Time Frame: Cycle 5 Day 1 (pre-dose) (1 cycle= 28 days)
Population: PK parameter analysis set was subset of safety analysis set (participants who received at least 1 dose of study drug) with participants who had at least 1 of PK parameters of interest for measured analytes related to study drug (i.e., sasanlimab). Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg)
Number analyzed (Participants) | 3 | 2
Microgram per milliliter | 37.97 (20) | 40.24 (NA) — Geometric coefficient of variation could not be calculated as at least 3 values were required and this criterion could not be fulfilled due to lack of available data.

24. Secondary Outcome: Phase 2 of Sub-Study A: Pre-dose Concentration During Multiple Dosing (Ctrough) of Sasanlimab
Time Frame: Cycle 5 Day 1 (pre-dose) (1 cycle= 28 days)
Population: as for outcome 2
Arm/Group | Phase 2: Sasanlimab + Encorafenib + Binimetinib
Number analyzed (Participants) | 0

25. Secondary Outcome: Phase 1b of Sub-Study A: Ctrough of Encorafenib
Time Frame: Day 1 (pre-dose) of Cycle 1, 2 and 5; Day 15 of Cycle 1 (1 cycle= 28 days)
Population: PK parameter analysis set was subset of safety analysis set (participants who received at least 1 dose of study drug) with participants who had at least 1 of PK parameters of interest for measured analytes related to study drug. Here, 'Number Analyzed' signifies participants evaluable at specified timepoints. For 'Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg)' arm, samples were not analyzed for Cycle 2 Day 1 as it was collected incorrectly due to time deviation for visits.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg)
Number analyzed (Participants) | 4 | 9
Nanograms per milliliter
  Cycle 1 Day 1 | NA (NA) — Data could not be calculated as values were below lower limit of quantification. | NA (NA) — Data could not be calculated as values were below lower limit of quantification.
  Cycle 1 Day 15: number analyzed (Participants) | 2 | 4
  Cycle 1 Day 15 | 12.2 (176) | 18.5 (50)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 4
  Cycle 2 Day 1 |  | 11.1 (204)
  Cycle 5 Day 1: number analyzed (Participants) | 1 | 2
  Cycle 5 Day 1 | 5.0 (NA) — Geometric coefficient of variation could not be calculated for single participant | 7.8 (191)

26. Secondary Outcome: Phase 2 of Sub-Study A: Ctrough of Encorafenib
Time Frame: Cycle 5 Day 1 (pre-dose)
Population: as for outcome 2
Arm/Group | Phase 2: Sasanlimab + Encorafenib + Binimetinib
Number analyzed (Participants) | 0

27. Secondary Outcome: Phase 1b of Sub-Study A: Ctrough of Binimetinib
Time Frame: Day 1 (pre-dose) of Cycles 1, 2, and 5 (1 cycle= 28 days)
Population: PK parameter analysis set was subset of safety analysis set (participants who received at least 1 dose of study drug) with participants who had at least 1 of PK parameters of interest for measured analytes related to study drug. Here, 'Overall Number Analyzed' signifies participants evaluable for this outcome measure. Here, 'Number Analyzed' signifies participants evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg)
Number analyzed (Participants) | 1 | 4
Nanograms per milliliter
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0
  Cycle 2 Day 1 | 19.2 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 40.9 (98)
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 3
  Cycle 5 Day 1 |  | 35.7 (67)

28. Secondary Outcome: Phase 2 of Sub-Study A: Ctrough of Binimetinib
Time Frame: Cycle 5 Day 1 (pre-dose)
Population: as for outcome 2
Arm/Group | Phase 2: Sasanlimab + Encorafenib + Binimetinib
Number analyzed (Participants) | 0

29. Secondary Outcome: Phase 1b of Sub-Study A: Number of Participants With Positive Anti-Drug Antibody (ADA) and Neutralizing Antibody (NAb) Against Sasanlimab
Description: In this outcome measure, number of ADA-positive and NAb-positive participants has been presented. A participant was considered ADA (or NAb) positive if (1) baseline titer was missing or negative and participant had >= 1 post-treatment positive titer (treatment-induced), or (2) positive titer at baseline and had a >= [4-fold dilution increase] in titer (equivalent to 0.602 unit increase in logarithm to base 10 (log10) titer from baseline in >= 1 post-treatment sample (treatment-boosted).
Time Frame: Pre-dose on Cycle 1 Day 1 until end of treatment (up to approximately 255 days) (1 cycle= 28 days)
Population: Immunogenicity analysis set was a subset of the safety analysis set (participants who received at least 1 dose of study drug) and included participants who had at least 1 analyzed sasanlimab ADA/NAb sample. All participants included in 'Overall Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, 'Number Analyzed' signifies participants evaluated for ADA and NAb respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg)
Number analyzed (Participants) | 4 | 9
Participants
  ADA: number analyzed (Participants) | 4 | 7
  ADA | 0 | 1
  NAb: number analyzed (Participants) | 4 | 6
  NAb | 0 | 0

30. Secondary Outcome: Phase 2 of Sub-Study A: Number of Participants With Positive Anti-Drug Antibody (ADA) and Neutralizing Antibody (NAb) Against Sasanlimab
Time Frame: Pre-dose on Cycle 1 Day 1 until end of treatment
Population: as for outcome 2
Arm/Group | Phase 2: Sasanlimab + Encorafenib + Binimetinib
Number analyzed (Participants) | 0

31. Secondary Outcome: Phase 2 of Sub-Study A: Objective Response (OR) Rate by Programmed Death Ligand-1 (PD-L1) Expression at Baseline
Description: OR rate is defined as percentage of participants with CR or PR according to RECIST v1.1 based on investigator assessment. CR=complete disappearance of all target lesions with exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). PR=greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. OR by PD-L1 expression at baseline was planned to be assessed.
Time Frame: as for outcome 2
Population: as for outcome 2
Arm/Group | Phase 2: Sasanlimab + Encorafenib + Binimetinib
Number analyzed (Participants) | 0

32. Secondary Outcome: Phase 2 of Sub-Study A: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (EORTC QLQ-C30) Score
Description: EORTC QLQ-C30: consisted of 30 questions grouped into 5 functional scales (physical, role, cognitive, emotional, and social); a global health status/global quality of life scale; 3 symptom scales (fatigue, pain, nausea and vomiting); and 6 single items that assessed additional symptoms (dyspnea, appetite loss, sleep disturbance, constipation, and diarrhea), and financial impact. All scales and single item measures ranged in score from 0 to 100. Higher scores on the global health status/quality of life scale represent higher health status/quality of life. Higher scores on the functional scales represent higher levels of functioning. Higher scores on the symptom scales and single items represent a greater presence of symptoms or financial impact.
Time Frame: Baseline up to end of treatment
Population: Due to a business decision, no participant was enrolled in Phase 2 of sub-study A. Hence, Phase 2 was not initiated and there was no data collection for it.
Arm/Group | Phase 2: Sasanlimab + Encorafenib + Binimetinib
Number analyzed (Participants) | 0

33. Secondary Outcome: Phase 2 of Sub-Study A: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC), Quality of Life Questionnaire-Lung Cancer 13 (QLQ- LC13) Score
Description: The EORTC QLQ-LC13 is the lung cancer specific module of the EORTC Quality of Life Questionnaire. The EORTC QLQ-LC13 consisted of 13 questions which included 1 multi-item scale and 9 single items assessing symptoms (dyspnea, cough, hemoptysis, and site specific pain), side effects (sore mouth, dysphagia, peripheral neuropathy, and alopecia), and pain medication use. The item scale ranged from 1 to 4 (1 = Not at all; 4 = Very Much) where the EORTC-QLQ-LC13 scoring algorithm was applied to convert to a 0 to 100 point scale where 100 is best quality of life (QOL), for comparability. Higher scores are reflective of a greater presence of symptoms.
Time Frame: Baseline up to end of treatment
Population: as for outcome 32
Arm/Group | Phase 2: Sasanlimab + Encorafenib + Binimetinib
Number analyzed (Participants) | 0

34. Secondary Outcome: Phase 1b of Sub-Study B: Number of Participants With Adverse Events Graded According to NCI-CTCAE Version 5.0
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. AEs were graded by the investigator according to NCI CTCAE version 5.0; where Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life-threatening and Grade 5=death.
Time Frame: as for outcome 5
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg)
Number analyzed (Participants) | 3 | 6
Participants
  Grade 1 | 0 | 0
  Grade 2 | 1 | 0
  Grade 3 | 2 | 4
  Grade 4 | 0 | 1
  Grade 5 | 0 | 1

35. Secondary Outcome: Phase 2 of Sub-Study B: Number of Participants With Adverse Events Graded According to NCI-CTCAE Version 5.0
Description: as for outcome 34
Time Frame: as for outcome 5
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
Number analyzed (Participants) | 3 | 2 | 7
Participants
  Grade 1 | 0 | 0 | 1
  Grade 2 | 0 | 0 | 2
  Grade 3 | 2 | 2 | 2
  Grade 4 | 1 | 0 | 2
  Grade 5 | 0 | 0 | 0

36. Secondary Outcome: Phase 1b of Sub-Study B: Number of Participants With Shift From Baseline in Hematology Parameters Values Based on CTCAE V5.0
Description: Hematology parameters included: anemia, hemoglobin increased, leukocytosis, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased, white blood cell decreased. Laboratory abnormalities were graded as per NCI- CTCAE v 5.0 where, grade(G) 0= non-missing lab value that does not meet either of G1 through 4 criteria, G1=mild, G2=moderate, G3=severe and G4= life-threatening or disabling. Baseline is defined as the last assessment prior to the date/time of the first dose of study treatment. Number of participants with shift from baseline in hematology parameters by grades (as per CTCAE version 5.0) were reported.
Time Frame: From the start of study treatment (Cycle1 Day1) up to 30 days after last dose of study treatment (maximum exposure = 39.3 months; maximum follow-up approximately 39.66 months)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg)
Number analyzed (Participants) | 3 | 6
Participants
  Anemia: Grade 0 to 0 | 0 | 2
  Anemia: Grade 0 to 1 | 1 | 0
  Anemia: Grade 0 to 2 | 0 | 0
  Anemia: Grade 0 to 3 | 0 | 0
  Anemia: Grade 0 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 1 to 0 | 0 | 0
  Anemia: Grade 1 to 1 | 2 | 3
  Anemia: Grade 1 to 2 | 0 | 0
  Anemia: Grade 1 to 3 | 0 | 0
  Anemia: Grade 1 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 2 to 0 | 0 | 0
  Anemia: Grade 2 to 1 | 0 | 0
  Anemia: Grade 2 to 2 | 0 | 1
  Anemia: Grade 2 to 3 | 0 | 0
  Anemia: Grade 2 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 3 to 0 | 0 | 0
  Anemia: Grade 3 to 1 | 0 | 0
  Anemia: Grade 3 to 2 | 0 | 0
  Anemia: Grade 3 to 3 | 0 | 0
  Anemia: Grade 3 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 4 to 0 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 4 to 1 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 4 to 2 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 4 to 3 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 4 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Hemoglobin increased: Grade 0 to 0 | 3 | 6
  Hemoglobin increased: Grade 0 to 1 | 0 | 0
  Hemoglobin increased: Grade 0 to 2 | 0 | 0
  Hemoglobin increased: Grade 0 to 3 | 0 | 0
  Hemoglobin increased: Grade 0 to 4 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 1 to 0 | 0 | 0
  Hemoglobin increased: Grade 1 to 1 | 0 | 0
  Hemoglobin increased: Grade 1 to 2 | 0 | 0
  Hemoglobin increased: Grade 1 to 3 | 0 | 0
  Hemoglobin increased: Grade 1 to 4 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 2 to 0 | 0 | 0
  Hemoglobin increased: Grade 2 to 1 | 0 | 0
  Hemoglobin increased: Grade 2 to 2 | 0 | 0
  Hemoglobin increased: Grade 2 to 3 | 0 | 0
  Hemoglobin increased: Grade 2 to 4 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 3 to 0 | 0 | 0
  Hemoglobin increased: Grade 3 to 1 | 0 | 0
  Hemoglobin increased: Grade 3 to 2 | 0 | 0
  Hemoglobin increased: Grade 3 to 3 | 0 | 0
  Hemoglobin increased: Grade 3 to 4 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 4 to 0 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 4 to 1 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 4 to 2 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 4 to 3 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 4 to 4 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Leukocytosis: Grade 0 to 0 | 3 | 6
  Leukocytosis: Grade 0 to 1 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 0 to 2 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 0 to 3 | 0 | 0
  Leukocytosis: Grade 0 to 4 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 1 to 0 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 1 to 1 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 1 to 2 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 1 to 3 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 1 to 4 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 2 to 0 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 2 to 1 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 2 to 2 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 2 to 3 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 2 to 4 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 3 to 0 | 0 | 0
  Leukocytosis: Grade 3 to 1 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 3 to 2 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 3 to 3 | 0 | 0
  Leukocytosis: Grade 3 to 4 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 4 to 0 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 4 to 1 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 4 to 2 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 4 to 3 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 4 to 4 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Lymphocyte count decreased: Grade 0 to 0 | 1 | 1
  Lymphocyte count decreased: Grade 0 to 1 | 0 | 0
  Lymphocyte count decreased: Grade 0 to 2 | 0 | 1
  Lymphocyte count decreased: Grade 0 to 3 | 0 | 1
  Lymphocyte count decreased: Grade 0 to 4 | 0 | 1
  Lymphocyte count decreased: Grade 1 to 0 | 0 | 0
  Lymphocyte count decreased: Grade 1 to 1 | 0 | 0
  Lymphocyte count decreased: Grade 1 to 2 | 2 | 0
  Lymphocyte count decreased: Grade 1 to 3 | 0 | 0
  Lymphocyte count decreased: Grade 1 to 4 | 0 | 1
  Lymphocyte count decreased: Grade 2 to 0 | 0 | 0
  Lymphocyte count decreased: Grade 2 to 1 | 0 | 0
  Lymphocyte count decreased: Grade 2 to 2 | 0 | 1
  Lymphocyte count decreased: Grade 2 to 3 | 0 | 0
  Lymphocyte count decreased: Grade 2 to 4 | 0 | 0
  Lymphocyte count decreased: Grade 3 to 0 | 0 | 00
  Lymphocyte count decreased: Grade 3 to 1 | 0 | 0
  Lymphocyte count decreased: Grade 3 to 2 | 0 | 0
  Lymphocyte count decreased: Grade 3 to 3 | 0 | 0
  Lymphocyte count decreased: Grade 3 to 4 | 0 | 0
  Lymphocyte count decreased: Grade 4 to 0 | 0 | 0
  Lymphocyte count decreased: Grade 4 to 1 | 0 | 0
  Lymphocyte count decreased: Grade 4 to 2 | 0 | 0
  Lymphocyte count decreased: Grade 4 to 3 | 0 | 0
  Lymphocyte count decreased: Grade 4 to 4 | 0 | 0
  Lymphocyte count increased: Grade 0 to 0 | 3 | 6
  Lymphocyte count increased: Grade 0 to 1 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 0 to 2 | 0 | 0
  Lymphocyte count increased: Grade 0 to 3 | 0 | 0
  Lymphocyte count increased: Grade 0 to 4 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 1 to 0 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 1 to 1 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 1 to 2 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 1 to 3 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 1 to 4 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 2 to 0 | 0 | 0
  Lymphocyte count increased: Grade 2 to 1 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 2 to 2 | 0 | 0
  Lymphocyte count increased: Grade 2 to 3 | 0 | 0
  Lymphocyte count increased: Grade 2 to 4 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 3 to 0 | 0 | 0
  Lymphocyte count increased: Grade 3 to 1 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 3 to 2 | 0 | 0
  Lymphocyte count increased: Grade 3 to 3 | 0 | 0
  Lymphocyte count increased: Grade 3 to 4 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 4 to 0 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 4 to 1 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 4 to 2 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 4 to 3 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 4 to 4 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Neutrophil count decreased: Grade 0 to 0 | 3 | 6
  Neutrophil count decreased: Grade 0 to 1 | 0 | 0
  Neutrophil count decreased: Grade 0 to 2 | 0 | 0
  Neutrophil count decreased: Grade 0 to 3 | 0 | 0
  Neutrophil count decreased: Grade 0 to 4 | 0 | 0
  Neutrophil count decreased: Grade 1 to 0 | 0 | 0
  Neutrophil count decreased: Grade 1 to 1 | 0 | 0
  Neutrophil count decreased: Grade 1 to 2 | 0 | 0
  Neutrophil count decreased: Grade 1 to 3 | 0 | 0
  Neutrophil count decreased: Grade 1 to 4 | 0 | 0
  Neutrophil count decreased: Grade 2 to 0 | 0 | 0
  Neutrophil count decreased: Grade 2 to 1 | 0 | 0
  Neutrophil count decreased: Grade 2 to 2 | 0 | 0
  Neutrophil count decreased: Grade 2 to 3 | 0 | 0
  Neutrophil count decreased: Grade 2 to 4 | 0 | 0
  Neutrophil count decreased: Grade 3 to 0 | 0 | 0
  Neutrophil count decreased: Grade 3 to 1 | 0 | 0
  Neutrophil count decreased: Grade 3 to 2 | 0 | 0
  Neutrophil count decreased: Grade 3 to 3 | 0 | 0
  Neutrophil count decreased: Grade 3 to 4 | 0 | 0
  Neutrophil count decreased: Grade 4 to 0 | 0 | 0
  Neutrophil count decreased: Grade 4 to 1 | 0 | 0
  Neutrophil count decreased: Grade 4 to 2 | 0 | 0
  Neutrophil count decreased: Grade 4 to 3 | 0 | 0
  Neutrophil count decreased: Grade 4 to 4 | 0 | 0
  Platelet count decreased: Grade 0 to 0 | 2 | 5
  Platelet count decreased: Grade 0 to 1 | 1 | 1
  Platelet count decreased: Grade 0 to 2 | 0 | 0
  Platelet count decreased: Grade 0 to 3 | 0 | 0
  Platelet count decreased: Grade 0 to 4 | 0 | 0
  Platelet count decreased: Grade 1 to 0 | 0 | 0
  Platelet count decreased: Grade 1 to 1 | 0 | 0
  Platelet count decreased: Grade 1 to 2 | 0 | 0
  Platelet count decreased: Grade 1 to 3 | 0 | 0
  Platelet count decreased: Grade 1 to 4 | 0 | 0
  Platelet count decreased: Grade 2 to 0 | 0 | 0
  Platelet count decreased: Grade 2 to 1 | 0 | 0
  Platelet count decreased: Grade 2 to 2 | 0 | 0
  Platelet count decreased: Grade 2 to 3 | 0 | 0
  Platelet count decreased: Grade 2 to 4 | 0 | 0
  Platelet count decreased: Grade 3 to 0 | 0 | 0
  Platelet count decreased: Grade 3 to 1 | 0 | 0
  Platelet count decreased: Grade 3 to 2 | 0 | 0
  Platelet count decreased: Grade 3 to 3 | 0 | 0
  Platelet count decreased: Grade 3 to 4 | 0 | 0
  Platelet count decreased: Grade 4 to 0 | 0 | 0
  Platelet count decreased: Grade 4 to 1 | 0 | 0
  Platelet count decreased: Grade 4 to 2 | 0 | 0
  Platelet count decreased: Grade 4 to 3 | 0 | 0
  Platelet count decreased: Grade 4 to 4 | 0 | 0
  White blood cell decreased: Grade 0 to 0 | 3 | 5
  White blood cell decreased: Grade 0 to 1 | 0 | 1
  White blood cell decreased: Grade 0 to 2 | 0 | 0
  White blood cell decreased: Grade 0 to 3 | 0 | 0
  White blood cell decreased: Grade 0 to 4 | 0 | 0
  White blood cell decreased: Grade 1 to 0 | 0 | 0
  White blood cell decreased: Grade 1 to 1 | 0 | 0
  White blood cell decreased: Grade 1 to 2 | 0 | 0
  White blood cell decreased: Grade 1 to 3 | 0 | 0
  White blood cell decreased: Grade 1 to 4 | 0 | 0
  White blood cell decreased: Grade 2 to 0 | 0 | 0
  White blood cell decreased: Grade 2 to 1 | 0 | 0
  White blood cell decreased: Grade 2 to 2 | 0 | 0
  White blood cell decreased: Grade 2 to 3 | 0 | 0
  White blood cell decreased: Grade 2 to 4 | 0 | 0
  White blood cell decreased: Grade 3 to 0 | 0 | 0
  White blood cell decreased: Grade 3 to 1 | 0 | 0
  White blood cell decreased: Grade 3 to 2 | 0 | 0
  White blood cell decreased: Grade 3 to 3 | 0 | 0
  White blood cell decreased: Grade 3 to 4 | 0 | 0
  White blood cell decreased: Grade 4 to 0 | 0 | 0
  White blood cell decreased: Grade 4 to 1 | 0 | 0
  White blood cell decreased: Grade 4 to 2 | 0 | 0
  White blood cell decreased: Grade 4 to 3 | 0 | 0
  White blood cell decreased: Grade 4 to 4 | 0 | 0

37. Secondary Outcome: Phase 1b of Sub-Study B: Number of Participants With Shift From Baseline in Chemistry Parameters Values Based on CTCAE V5.0
Description: Chemistry parameters included: alanine aminotransferase (ALT) increased, alkaline phosphatase (ALP) increased, aspartate aminotransferase (AST) increased, blood bilirubin increased, creatinine phosphokinase (CPK) increased, chronic kidney disease (CKD), creatinine increased, hypercalcemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, hyponatremia, lipase increased, serum amylase increased. Chemistry abnormalities were graded as per NCI- CTCAE v 5.0 where, grade(G) 0= non-missing lab value that does not meet either of G1 through 4 criteria, G1=mild, G2=moderate, G3=severe and G4= life-threatening or disabling. Baseline is defined as the last assessment prior to the date/time of the first dose of study treatment. Number of participants with shift from baseline in hematology parameters by grades (as per CTCAE version 5.0) were reported.
Time Frame: as for outcome 5
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg)
Number analyzed (Participants) | 3 | 6
Participants
  ALT increased: Grade 0 to 0 | 1 | 5
  ALT increased: Grade 0 to 1 | 2 | 0
  ALT increased: Grade 0 to 2 | 0 | 1
  ALT increased: Grade 0 to 3 | 0 | 0
  ALT increased: Grade 0 to 4 | 0 | 0
  ALT increased: Grade 1 to 0 | 0 | 0
  ALT increased: Grade 1 to 1 | 0 | 0
  ALT increased: Grade 1 to 2 | 0 | 0
  ALT increased: Grade 1 to 3 | 0 | 0
  ALT increased: Grade 1 to 4 | 0 | 0
  ALT increased: Grade 2 to 0 | 0 | 0
  ALT increased: Grade 2 to 1 | 0 | 0
  ALT increased: Grade 2 to 2 | 0 | 0
  ALT increased: Grade 2 to 3 | 0 | 0
  ALT increased: Grade 2 to 4 | 0 | 0
  ALT increased: Grade 3 to 0 | 0 | 0
  ALT increased: Grade 3 to 1 | 0 | 0
  ALT increased: Grade 3 to 2 | 0 | 0
  ALT increased: Grade 3 to 3 | 0 | 0
  ALT increased: Grade 3 to 4 | 0 | 0
  ALT increased: Grade 4 to 0 | 0 | 0
  ALT increased: Grade 4 to 1 | 0 | 0
  ALT increased: Grade 4 to 2 | 0 | 0
  ALT increased: Grade 4 to 3 | 0 | 0
  ALT increased: Grade 4 to 4 | 0 | 0
  ALP increased: Grade 0 to 0 | 2 | 4
  ALP increased: Grade 0 to 1 | 0 | 2
  ALP increased: Grade 0 to 2 | 0 | 0
  ALP increased: Grade 0 to 3 | 0 | 0
  ALP increased: Grade 0 to 4 | 0 | 0
  ALP increased: Grade 1 to 0 | 0 | 0
  ALP increased: Grade 1 to 1 | 0 | 0
  ALP increased: Grade 1 to 2 | 1 | 0
  ALP increased: Grade 1 to 3 | 0 | 0
  ALP increased: Grade 1 to 4 | 0 | 0
  ALP increased: Grade 2 to 0 | 0 | 0
  ALP increased: Grade 2 to 1 | 0 | 0
  ALP increased: Grade 2 to 2 | 0 | 0
  ALP increased: Grade 2 to 3 | 0 | 0
  ALP increased: Grade 2 to 4 | 0 | 0
  ALP increased: Grade 3 to 0 | 0 | 0
  ALP increased: Grade 3 to 1 | 0 | 0
  ALP increased: Grade 3 to 2 | 0 | 0
  ALP increased: Grade 3 to 3 | 0 | 0
  ALP increased: Grade 3 to 4 | 0 | 0
  ALP increased: Grade 4 to 0 | 0 | 0
  ALP increased: Grade 4 to 1 | 0 | 0
  ALP increased: Grade 4 to 2 | 0 | 0
  ALP increased: Grade 4 to 3 | 0 | 0
  ALP increased: Grade 4 to 4 | 0 | 0
  AST increased: Grade 0 to 0 | 0 | 5
  AST increased: Grade 0 to 1 | 1 | 0
  AST increased: Grade 0 to 2 | 0 | 0
  AST increased: Grade 0 to 3 | 0 | 1
  AST increased: Grade 0 to 4 | 0 | 0
  AST increased: Grade 1 to 0 | 1 | 0
  AST increased: Grade 1 to 1 | 1 | 0
  AST increased: Grade 1 to 2 | 0 | 0
  AST increased: Grade 1 to 3 | 0 | 0
  AST increased: Grade 1 to 4 | 0 | 0
  AST increased: Grade 2 to 0 | 0 | 0
  AST increased: Grade 2 to 1 | 0 | 0
  AST increased: Grade 2 to 2 | 0 | 0
  AST increased: Grade 2 to 3 | 0 | 0
  AST increased: Grade 2 to 4 | 0 | 0
  AST increased: Grade 3 to 0 | 0 | 0
  AST increased: Grade 3 to 1 | 0 | 0
  AST increased: Grade 3 to 2 | 0 | 0
  AST increased: Grade 3 to 3 | 0 | 0
  AST increased: Grade 3 to 4 | 0 | 0
  AST increased: Grade 4 to 0 | 0 | 0
  AST increased: Grade 4 to 1 | 0 | 0
  AST increased: Grade 4 to 2 | 0 | 0
  AST increased: Grade 4 to 3 | 0 | 0
  AST increased: Grade 4 to 4 | 0 | 0
  Blood bilirubin increased: Grade 0 to 0 | 3 | 6
  Blood bilirubin increased: Grade 0 to 1 | 0 | 0
  Blood bilirubin increased: Grade 0 to 2 | 0 | 0
  Blood bilirubin increased: Grade 0 to 3 | 0 | 0
  Blood bilirubin increased: Grade 0 to 4 | 0 | 0
  Blood bilirubin increased: Grade 1 to 0 | 0 | 0
  Blood bilirubin increased: Grade 1 to 1 | 0 | 0
  Blood bilirubin increased: Grade 1 to 2 | 0 | 0
  Blood bilirubin increased: Grade 1 to 3 | 0 | 0
  Blood bilirubin increased: Grade 1 to 4 | 0 | 0
  Blood bilirubin increased: Grade 2 to 0 | 0 | 0
  Blood bilirubin increased: Grade 2 to 1 | 0 | 0
  Blood bilirubin increased: Grade 2 to 2 | 0 | 0
  Blood bilirubin increased: Grade 2 to 3 | 0 | 0
  Blood bilirubin increased: Grade 2 to 4 | 0 | 0
  Blood bilirubin increased: Grade 3 to 0 | 0 | 0
  Blood bilirubin increased: Grade 3 to 1 | 0 | 0
  Blood bilirubin increased: Grade 3 to 2 | 0 | 0
  Blood bilirubin increased: Grade 3 to 3 | 0 | 0
  Blood bilirubin increased: Grade 3 to 4 | 0 | 0
  Blood bilirubin increased: Grade 4 to 0 | 0 | 0
  Blood bilirubin increased: Grade 4 to 1 | 0 | 0
  Blood bilirubin increased: Grade 4 to 2 | 0 | 0
  Blood bilirubin increased: Grade 4 to 3 | 0 | 0
  Blood bilirubin increased: Grade 4 to 4 | 0 | 0
  CPK increased: Grade 0 to 0 | 3 | 5
  CPK increased: Grade 0 to 1 | 0 | 0
  CPK increased: Grade 0 to 2 | 0 | 0
  CPK increased: Grade 0 to 3 | 0 | 0
  CPK increased: Grade 0 to 4 | 0 | 0
  CPK increased: Grade 1 to 0 | 0 | 1
  CPK increased: Grade 1 to 1 | 0 | 0
  CPK increased: Grade 1 to 2 | 0 | 0
  CPK increased: Grade 1 to 3 | 0 | 0
  CPK increased: Grade 1 to 4 | 0 | 0
  CPK increased: Grade 2 to 0 | 0 | 0
  CPK increased: Grade 2 to 1 | 0 | 0
  CPK increased: Grade 2 to 2 | 0 | 0
  CPK increased: Grade 2 to 3 | 0 | 0
  CPK increased: Grade 2 to 4 | 0 | 0
  CPK increased: Grade 3 to 0 | 0 | 0
  CPK increased: Grade 3 to 1 | 0 | 0
  CPK increased: Grade 3 to 2 | 0 | 0
  CPK increased: Grade 3 to 3 | 0 | 0
  CPK increased: Grade 3 to 4 | 0 | 0
  CPK increased: Grade 4 to 0 | 0 | 0
  CPK increased: Grade 4 to 1 | 0 | 0
  CPK increased: Grade 4 to 2 | 0 | 0
  CPK increased: Grade 4 to 3 | 0 | 0
  CPK increased: Grade 4 to 4 | 0 | 0
  Chronic kidney disease: Grade 0 to 0 | 1 | 0
  Chronic kidney disease: Grade 0 to 1 | 1 | 2
  Chronic kidney disease: Grade 0 to 2 | 0 | 1
  Chronic kidney disease: Grade 0 to 3 | 0 | 0
  Chronic kidney disease: Grade 0 to 4 | 0 | 0
  Chronic kidney disease: Grade 1 to 0 | 0 | 0
  Chronic kidney disease: Grade 1 to 1 | 0 | 0
  Chronic kidney disease: Grade 1 to 2 | 00 | 1
  Chronic kidney disease: Grade 1 to 3 | 0 | 0
  Chronic kidney disease: Grade 1 to 4 | 0 | 0
  Chronic kidney disease: Grade 2 to 0 | 0 | 0
  Chronic kidney disease: Grade 2 to 1 | 0 | 0
  Chronic kidney disease: Grade 2 to 2 | 1 | 2
  Chronic kidney disease: Grade 2 to 3 | 0 | 0
  Chronic kidney disease: Grade 2 to 4 | 0 | 0
  Chronic kidney disease: Grade 3 to 0 | 0 | 0
  Chronic kidney disease: Grade 3 to 1 | 0 | 0
  Chronic kidney disease: Grade 3 to 2 | 0 | 0
  Chronic kidney disease: Grade 3 to 3 | 0 | 0
  Chronic kidney disease: Grade 3 to 4 | 0 | 0
  Chronic kidney disease: Grade 4 to 0 | 0 | 0
  Chronic kidney disease: Grade 4 to 1 | 0 | 0
  Chronic kidney disease: Grade 4 to 2 | 0 | 0
  Chronic kidney disease: Grade 4 to 3 | 0 | 0
  Chronic kidney disease: Grade 4 to 4 | 0 | 0
  Creatinine increased: Grade 0 to 0 | 2 | 3
  Creatinine increased: Grade 0 to 1 | 0 | 0
  Creatinine increased: Grade 0 to 2 | 0 | 0
  Creatinine increased: Grade 0 to 3 | 0 | 0
  Creatinine increased: Grade 0 to 4 | 0 | 0
  Creatinine increased: Grade 1 to 0 | 0 | 0
  Creatinine increased: Grade 1 to 1 | 1 | 2
  Creatinine increased: Grade 1 to 2 | 0 | 1
  Creatinine increased: Grade 1 to 3 | 0 | 0
  Creatinine increased: Grade 1 to 4 | 0 | 0
  Creatinine increased: Grade 2 to 0 | 0 | 0
  Creatinine increased: Grade 2 to 1 | 0 | 0
  Creatinine increased: Grade 2 to 2 | 0 | 0
  Creatinine increased: Grade 2 to 3 | 0 | 0
  Creatinine increased: Grade 2 to 4 | 0 | 0
  Creatinine increased: Grade 3 to 0 | 0 | 0
  Creatinine increased: Grade 3 to 1 | 0 | 0
  Creatinine increased: Grade 3 to 2 | 0 | 0
  Creatinine increased: Grade 3 to 3 | 0 | 0
  Creatinine increased: Grade 3 to 4 | 0 | 0
  Creatinine increased: Grade 4 to 0 | 0 | 0
  Creatinine increased: Grade 4 to 1 | 0 | 0
  Creatinine increased: Grade 4 to 2 | 0 | 0
  Creatinine increased: Grade 4 to 3 | 0 | 0
  Creatinine increased: Grade 4 to 4 | 0 | 0
  Hypercalcemia: Grade 0 to 0 | 1 | 5
  Hypercalcemia: Grade 0 to 1 | 2 | 1
  Hypercalcemia: Grade 0 to 2 | 0 | 0
  Hypercalcemia: Grade 0 to 3 | 0 | 0
  Hypercalcemia: Grade 0 to 4 | 0 | 0
  Hypercalcemia: Grade 1 to 0 | 0 | 0
  Hypercalcemia: Grade 1 to 1 | 0 | 0
  Hypercalcemia: Grade 1 to 2 | 0 | 0
  Hypercalcemia: Grade 1 to 3 | 0 | 0
  Hypercalcemia: Grade 1 to 4 | 0 | 0
  Hypercalcemia: Grade 2 to 0 | 0 | 0
  Hypercalcemia: Grade 2 to 1 | 0 | 0
  Hypercalcemia: Grade 2 to 2 | 0 | 0
  Hypercalcemia: Grade 2 to 3 | 0 | 0
  Hypercalcemia: Grade 2 to 4 | 0 | 0
  Hypercalcemia: Grade 3 to 0 | 0 | 0
  Hypercalcemia: Grade 3 to 1 | 0 | 0
  Hypercalcemia: Grade 3 to 2 | 0 | 0
  Hypercalcemia: Grade 3 to 3 | 0 | 0
  Hypercalcemia: Grade 3 to 4 | 0 | 0
  Hypercalcemia: Grade 4 to 0 | 0 | 0
  Hypercalcemia: Grade 4 to 1 | 0 | 0
  Hypercalcemia: Grade 4 to 2 | 0 | 0
  Hypercalcemia: Grade 4 to 3 | 0 | 0
  Hypercalcemia: Grade 4 to 4 | 0 | 0
  Hyperkalemia: Grade 0 to 0 | 2 | 5
  Hyperkalemia: Grade 0 to 1 | 1 | 1
  Hyperkalemia: Grade 0 to 2 | 0 | 0
  Hyperkalemia: Grade 0 to 3 | 0 | 0
  Hyperkalemia: Grade 0 to 4 | 0 | 0
  Hyperkalemia: Grade 1 to 0 | 0 | 0
  Hyperkalemia: Grade 1 to 1 | 0 | 0
  Hyperkalemia: Grade 1 to 2 | 0 | 0
  Hyperkalemia: Grade 1 to 3 | 0 | 0
  Hyperkalemia: Grade 1 to 4 | 0 | 0
  Hyperkalemia: Grade 2 to 0 | 0 | 0
  Hyperkalemia: Grade 2 to 1 | 0 | 0
  Hyperkalemia: Grade 2 to 2 | 0 | 0
  Hyperkalemia: Grade 2 to 3 | 0 | 0
  Hyperkalemia: Grade 2 to 4 | 0 | 0
  Hyperkalemia: Grade 3 to 0 | 0 | 0
  Hyperkalemia: Grade 3 to 1 | 0 | 0
  Hyperkalemia: Grade 3 to 2 | 0 | 0
  Hyperkalemia: Grade 3 to 3 | 0 | 0
  Hyperkalemia: Grade 3 to 4 | 0 | 0
  Hyperkalemia: Grade 4 to 0 | 0 | 0
  Hyperkalemia: Grade 4 to 1 | 0 | 0
  Hyperkalemia: Grade 4 to 2 | 0 | 0
  Hyperkalemia: Grade 4 to 3 | 0 | 0
  Hyperkalemia: Grade 4 to 4 | 0 | 0
  Hypermagnesemia: Grade 0 to 0 | 3 | 6
  Hypermagnesemia: Grade 0 to 1 | 0 | 0
  Hypermagnesemia: Grade 0 to 2 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 0 to 3 | 0 | 0
  Hypermagnesemia: Grade 0 to 4 | 0 | 0
  Hypermagnesemia: Grade 1 to 0 | 0 | 0
  Hypermagnesemia: Grade 1 to 1 | 0 | 0
  Hypermagnesemia: Grade 1 to 2 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 1 to 3 | 0 | 0
  Hypermagnesemia: Grade 1 to 4 | 0 | 0
  Hypermagnesemia: Grade 2 to 0 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 2 to 1 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 2 to 2 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 2 to 3 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 2 to 4 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 3 to 0 | 0 | 0
  Hypermagnesemia: Grade 3 to 1 | 0 | 0
  Hypermagnesemia: Grade 3 to 2 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 3 to 3 | 0 | 0
  Hypermagnesemia: Grade 3 to 4 | 0 | 0
  Hypermagnesemia: Grade 4 to 0 | 0 | 0
  Hypermagnesemia: Grade 4 to 1 | 0 | 0
  Hypermagnesemia: Grade 4 to 2 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 4 to 3 | 0 | 0
  Hypermagnesemia: Grade 4 to 4 | 0 | 0
  Hypernatremia: Grade 0 to 0 | 3 | 6
  Hypernatremia: Grade 0 to 1 | 0 | 0
  Hypernatremia: Grade 0 to 2 | 0 | 0
  Hypernatremia: Grade 0 to 3 | 0 | 0
  Hypernatremia: Grade 0 to 4 | 0 | 0
  Hypernatremia: Grade 1 to 0 | 0 | 0
  Hypernatremia: Grade 1 to 1 | 0 | 0
  Hypernatremia: Grade 1 to 2 | 0 | 0
  Hypernatremia: Grade 1 to 3 | 0 | 0
  Hypernatremia: Grade 1 to 4 | 0 | 0
  Hypernatremia: Grade 2 to 0 | 0 | 0
  Hypernatremia: Grade 2 to 1 | 0 | 0
  Hypernatremia: Grade 2 to 2 | 0 | 0
  Hypernatremia: Grade 2 to 3 | 0 | 0
  Hypernatremia: Grade 2 to 4 | 0 | 0
  Hypernatremia: Grade 3 to 0 | 0 | 0
  Hypernatremia: Grade 3 to 1 | 0 | 0
  Hypernatremia: Grade 3 to 2 | 0 | 0
  Hypernatremia: Grade 3 to 3 | 0 | 0
  Hypernatremia: Grade 3 to 4 | 0 | 0
  Hypernatremia: Grade 4 to 0 | 0 | 0
  Hypernatremia: Grade 4 to 1 | 0 | 0
  Hypernatremia: Grade 4 to 2 | 0 | 0
  Hypernatremia: Grade 4 to 3 | 0 | 0
  Hypernatremia: Grade 4 to 4 | 0 | 0
  Hypoalbuminemia: Grade 0 to 0 | 2 | 2
  Hypoalbuminemia: Grade 0 to 1 | 1 | 1
  Hypoalbuminemia: Grade 0 to 2 | 0 | 1
  Hypoalbuminemia: Grade 0 to 3 | 0 | 0
  Hypoalbuminemia: Grade 0 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 1 to 0 | 0 | 0
  Hypoalbuminemia: Grade 1 to 1 | 0 | 0
  Hypoalbuminemia: Grade 1 to 2 | 0 | 1
  Hypoalbuminemia: Grade 1 to 3 | 0 | 0
  Hypoalbuminemia: Grade 1 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 2 to 0 | 0 | 0
  Hypoalbuminemia: Grade 2 to 1 | 0 | 0
  Hypoalbuminemia: Grade 2 to 2 | 0 | 1
  Hypoalbuminemia: Grade 2 to 3 | 0 | 0
  Hypoalbuminemia: Grade 2 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 3 to 0 | 0 | 0
  Hypoalbuminemia: Grade 3 to 1 | 0 | 0
  Hypoalbuminemia: Grade 3 to 2 | 0 | 0
  Hypoalbuminemia: Grade 3 to 3 | 0 | 0
  Hypoalbuminemia: Grade 3 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 4 to 0 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 4 to 1 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 4 to 2 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 4 to 3 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 4 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypocalcemia: Grade 0 to 0 | 3 | 6
  Hypocalcemia: Grade 0 to 1 | 0 | 0
  Hypocalcemia: Grade 0 to 2 | 0 | 0
  Hypocalcemia: Grade 0 to 3 | 0 | 0
  Hypocalcemia: Grade 0 to 4 | 0 | 0
  Hypocalcemia: Grade 1 to 0 | 0 | 0
  Hypocalcemia: Grade 1 to 1 | 0 | 0
  Hypocalcemia: Grade 1 to 2 | 0 | 0
  Hypocalcemia: Grade 1 to 3 | 0 | 0
  Hypocalcemia: Grade 1 to 4 | 0 | 0
  Hypocalcemia: Grade 2 to 0 | 0 | 0
  Hypocalcemia: Grade 2 to 1 | 0 | 0
  Hypocalcemia: Grade 2 to 2 | 0 | 0
  Hypocalcemia: Grade 2 to 3 | 0 | 0
  Hypocalcemia: Grade 2 to 4 | 0 | 0
  Hypocalcemia: Grade 3 to 0 | 0 | 0
  Hypocalcemia: Grade 3 to 1 | 0 | 0
  Hypocalcemia: Grade 3 to 2 | 0 | 0
  Hypocalcemia: Grade 3 to 3 | 0 | 0
  Hypocalcemia: Grade 3 to 4 | 0 | 0
  Hypocalcemia: Grade 4 to 0 | 0 | 0
  Hypocalcemia: Grade 4 to 1 | 0 | 0
  Hypocalcemia: Grade 4 to 2 | 0 | 0
  Hypocalcemia: Grade 4 to 3 | 0 | 0
  Hypocalcemia: Grade 4 to 4 | 0 | 0
  Hypoglycemia: Grade 0 to 0 | 2 | 5
  Hypoglycemia: Grade 0 to 1 | 1 | 1
  Hypoglycemia: Grade 0 to 2 | 0 | 0
  Hypoglycemia: Grade 0 to 3 | 0 | 0
  Hypoglycemia: Grade 0 to 4 | 0 | 0
  Hypoglycemia: Grade 1 to 0 | 0 | 0
  Hypoglycemia: Grade 1 to 1 | 0 | 0
  Hypoglycemia: Grade 1 to 2 | 0 | 0
  Hypoglycemia: Grade 1 to 3 | 0 | 0
  Hypoglycemia: Grade 1 to 4 | 0 | 0
  Hypoglycemia: Grade 2 to 0 | 0 | 0
  Hypoglycemia: Grade 2 to 1 | 0 | 0
  Hypoglycemia: Grade 2 to 2 | 0 | 0
  Hypoglycemia: Grade 2 to 3 | 0 | 0
  Hypoglycemia: Grade 2 to 4 | 0 | 0
  Hypoglycemia: Grade 3 to 0 | 0 | 0
  Hypoglycemia: Grade 3 to 1 | 0 | 0
  Hypoglycemia: Grade 3 to 2 | 0 | 0
  Hypoglycemia: Grade 3 to 3 | 0 | 0
  Hypoglycemia: Grade 3 to 4 | 0 | 0
  Hypoglycemia: Grade 4 to 0 | 0 | 0
  Hypoglycemia: Grade 4 to 1 | 0 | 0
  Hypoglycemia: Grade 4 to 2 | 0 | 0
  Hypoglycemia: Grade 4 to 3 | 0 | 0
  Hypoglycemia: Grade 4 to 4 | 0 | 0
  Hypokalemia: Grade 0 to 0 | 2 | 4
  Hypokalemia: Grade 0 to 1 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 0 to 2 | 1 | 2
  Hypokalemia: Grade 0 to 3 | 0 | 0
  Hypokalemia: Grade 0 to 4 | 0 | 0
  Hypokalemia: Grade 1 to 0 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 1 to 1 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 1 to 2 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 1 to 3 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 1 to 4 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 2 to 0 | 0 | 0
  Hypokalemia: Grade 2 to 1 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 2 to 2 | 0 | 0
  Hypokalemia: Grade 2 to 3 | 0 | 0
  Hypokalemia: Grade 2 to 4 | 0 | 0
  Hypokalemia: Grade 3 to 0 | 0 | 0
  Hypokalemia: Grade 3 to 1 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 3 to 2 | 0 | 0
  Hypokalemia: Grade 3 to 3 | 0 | 0
  Hypokalemia: Grade 3 to 4 | 0 | 0
  Hypokalemia: Grade 4 to 0 | 0 | 0
  Hypokalemia: Grade 4 to 1 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 4 to 2 | 0 | 0
  Hypokalemia: Grade 4 to 3 | 0 | 0
  Hypokalemia: Grade 4 to 4 | 0 | 0
  Hypomagnesemia: Grade 0 to 0 | 1 | 5
  Hypomagnesemia: Grade 0 to 1 | 1 | 1
  Hypomagnesemia: Grade 0 to 2 | 0 | 0
  Hypomagnesemia: Grade 0 to 3 | 0 | 0
  Hypomagnesemia: Grade 0 to 4 | 0 | 0
  Hypomagnesemia: Grade 1 to 0 | 0 | 0
  Hypomagnesemia: Grade 1 to 1 | 0 | 0
  Hypomagnesemia: Grade 1 to 2 | 0 | 0
  Hypomagnesemia: Grade 1 to 3 | 0 | 0
  Hypomagnesemia: Grade 1 to 4 | 0 | 0
  Hypomagnesemia: Grade 2 to 0 | 0 | 0
  Hypomagnesemia: Grade 2 to 1 | 1 | 0
  Hypomagnesemia: Grade 2 to 2 | 0 | 0
  Hypomagnesemia: Grade 2 to 3 | 0 | 0
  Hypomagnesemia: Grade 2 to 4 | 0 | 0
  Hypomagnesemia: Grade 3 to 0 | 0 | 0
  Hypomagnesemia: Grade 3 to 1 | 0 | 0
  Hypomagnesemia: Grade 3 to 2 | 0 | 0
  Hypomagnesemia: Grade 3 to 3 | 0 | 0
  Hypomagnesemia: Grade 3 to 4 | 0 | 0
  Hypomagnesemia: Grade 4 to 0 | 0 | 0
  Hypomagnesemia: Grade 4 to 1 | 0 | 0
  Hypomagnesemia: Grade 4 to 2 | 0 | 0
  Hypomagnesemia: Grade 4 to 3 | 0 | 0
  Hypomagnesemia: Grade 4 to 4 | 0 | 0
  Hyponatremia: Grade 0 to 0 | 2 | 4
  Hyponatremia: Grade 0 to 1 | 1 | 2
  Hyponatremia: Grade 0 to 2 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 0 to 3 | 0 | 0
  Hyponatremia: Grade 0 to 4 | 0 | 0
  Hyponatremia: Grade 1 to 0 | 0 | 0
  Hyponatremia: Grade 1 to 1 | 0 | 0
  Hyponatremia: Grade 1 to 2 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 1 to 3 | 0 | 0
  Hyponatremia: Grade 1 to 4 | 0 | 0
  Hyponatremia: Grade 2 to 0 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 2 to 1 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 2 to 2 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 2 to 3 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 2 to 4 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 3 to 0 | 0 | 0
  Hyponatremia: Grade 3 to 1 | 0 | 0
  Hyponatremia: Grade 3 to 2 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 3 to 3 | 0 | 0
  Hyponatremia: Grade 3 to 4 | 0 | 0
  Hyponatremia: Grade 4 to 0 | 0 | 0
  Hyponatremia: Grade 4 to 1 | 0 | 0
  Hyponatremia: Grade 4 to 2 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 4 to 3 | 0 | 0
  Hyponatremia: Grade 4 to 4 | 0 | 0
  Lipase increased: Grade 0 to 0 | 3 | 4
  Lipase increased: Grade 0 to 1 | 0 | 2
  Lipase increased: Grade 0 to 2 | 0 | 0
  Lipase increased: Grade 0 to 3 | 0 | 0
  Lipase increased: Grade 0 to 4 | 0 | 0
  Lipase increased: Grade 1 to 0 | 0 | 0
  Lipase increased: Grade 1 to 1 | 0 | 0
  Lipase increased: Grade 1 to 2 | 0 | 0
  Lipase increased: Grade 1 to 3 | 0 | 0
  Lipase increased: Grade 1 to 4 | 0 | 0
  Lipase increased: Grade 2 to 0 | 0 | 0
  Lipase increased: Grade 2 to 1 | 0 | 0
  Lipase increased: Grade 2 to 2 | 0 | 0
  Lipase increased: Grade 2 to 3 | 0 | 0
  Lipase increased: Grade 2 to 4 | 0 | 0
  Lipase increased: Grade 3 to 0 | 0 | 0
  Lipase increased: Grade 3 to 1 | 0 | 0
  Lipase increased: Grade 3 to 2 | 0 | 0
  Lipase increased: Grade 3 to 3 | 0 | 0
  Lipase increased: Grade 3 to 4 | 0 | 0
  Lipase increased: Grade 4 to 0 | 0 | 0
  Lipase increased: Grade 4 to 1 | 0 | 0
  Lipase increased: Grade 4 to 2 | 0 | 0
  Lipase increased: Grade 4 to 3 | 0 | 0
  Lipase increased: Grade 4 to 4 | 0 | 0
  Serum amylase increased: Grade 0 to 0 | 3 | 4
  Serum amylase increased: Grade 0 to 1 | 0 | 1
  Serum amylase increased: Grade 0 to 2 | 0 | 0
  Serum amylase increased: Grade 0 to 3 | 0 | 0
  Serum amylase increased: Grade 0 to 4 | 0 | 0
  Serum amylase increased: Grade 1 to 0 | 0 | 0
  Serum amylase increased: Grade 1 to 1 | 0 | 0
  Serum amylase increased: Grade 1 to 2 | 0 | 1
  Serum amylase increased: Grade 1 to 3 | 0 | 0
  Serum amylase increased: Grade 1 to 4 | 0 | 0
  Serum amylase increased: Grade 2 to 0 | 0 | 0
  Serum amylase increased: Grade 2 to 1 | 0 | 0
  Serum amylase increased: Grade 2 to 2 | 0 | 0
  Serum amylase increased: Grade 2 to 3 | 0 | 0
  Serum amylase increased: Grade 2 to 4 | 0 | 0
  Serum amylase increased: Grade 3 to 0 | 0 | 0
  Serum amylase increased: Grade 3 to 1 | 0 | 0
  Serum amylase increased: Grade 3 to 2 | 0 | 0
  Serum amylase increased: Grade 3 to 3 | 0 | 0
  Serum amylase increased: Grade 3 to 4 | 0 | 0
  Serum amylase increased: Grade 4 to 0 | 0 | 0
  Serum amylase increased: Grade 4 to 1 | 0 | 0
  Serum amylase increased: Grade 4 to 2 | 0 | 0
  Serum amylase increased: Grade 4 to 3 | 0 | 0
  Serum amylase increased: Grade 4 to 4 | 0 | 0

38. Secondary Outcome: Phase 2 of Sub-Study B: Number of Participants With Shift From Baseline in Hematology Parameter Values Based on CTCAE V5.0
Description: Hematology parameters included: anemia, hemoglobin increased, lymphocyte count decreased, leukocytosis, neutrophil count decreased, platelet count decreased, white blood cell decreased. Number of participants with shift from baseline in hematology parameters by grades as per CTCAE version 5.0 were reported. Grade 0= non-missing lab value that does not meet either of Grade 1 through 4 criteria; Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling.
Time Frame: as for outcome 5
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
Number analyzed (Participants) | 3 | 2 | 7
Participants
  Anemia: Grade 0 to 0 | 1 | 0 | 5
  Anemia: Grade 0 to 1 | 1 | 0 | 0
  Anemia: Grade 0 to 2 | 0 | 0 | 0
  Anemia: Grade 0 to 3 | 0 | 0 | 0
  Anemia: Grade 0 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 1 to 0 | 0 | 0 | 1
  Anemia: Grade 1 to 1 | 0 | 2 | 1
  Anemia: Grade 1 to 2 | 0 | 0 | 0
  Anemia: Grade 1 to 3 | 0 | 0 | 0
  Anemia: Grade 1 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 2 to 0 | 0 | 0 | 0
  Anemia: Grade 2 to 1 | 0 | 0 | 0
  Anemia: Grade 2 to 2 | 1 | 0 | 0
  Anemia: Grade 2 to 3 | 0 | 0 | 0
  Anemia: Grade 2 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 3 to 0 | 0 | 0 | 0
  Anemia: Grade 3 to 1 | 0 | 0 | 0
  Anemia: Grade 3 to 2 | 0 | 0 | 0
  Anemia: Grade 3 to 3 | 0 | 0 | 0
  Anemia: Grade 3 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 4 to 0 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 4 to 1 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 4 to 2 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 4 to 3 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Anemia: Grade 4 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for anemia.
  Hemoglobin increased: Grade 0 to 0 | 3 | 2 | 6
  Hemoglobin increased: Grade 0 to 1 | 0 | 0 | 1
  Hemoglobin increased: Grade 0 to 2 | 0 | 0 | 0
  Hemoglobin increased: Grade 0 to 3 | 0 | 0 | 0
  Hemoglobin increased: Grade 0 to 4 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 1 to 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 1 to 1 | 0 | 0 | 0
  Hemoglobin increased: Grade 1 to 2 | 0 | 0 | 0
  Hemoglobin increased: Grade 1 to 3 | 0 | 0 | 0
  Hemoglobin increased: Grade 1 to 4 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 2 to 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 2 to 1 | 0 | 0 | 0
  Hemoglobin increased: Grade 2 to 2 | 0 | 0 | 0
  Hemoglobin increased: Grade 2 to 3 | 0 | 0 | 0
  Hemoglobin increased: Grade 2 to 4 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 3 to 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 3 to 1 | 0 | 0 | 0
  Hemoglobin increased: Grade 3 to 2 | 0 | 0 | 0
  Hemoglobin increased: Grade 3 to 3 | 0 | 0 | 0
  Hemoglobin increased: Grade 3 to 4 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 4 to 0 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 4 to 1 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 4 to 2 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 4 to 3 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Hemoglobin increased: Grade 4 to 4 | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased. | NA — Grade 4 is not defined in CTCAE (i.e. Blank) therefore Grade 4 is NA for hemoglobin increased.
  Leukocytosis: Grade 0 to 0 | 3 | 2 | 7
  Leukocytosis: Grade 0 to 1 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 0 to 2 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 0 to 3 | 0 | 0 | 0
  Leukocytosis: Grade 0 to 4 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 1 to 0 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 1 to 1 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 1 to 2 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 1 to 3 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 1 to 4 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 2 to 0 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 2 to 1 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 2 to 2 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 2 to 3 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 2 to 4 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 3 to 0 | 0 | 0 | 0
  Leukocytosis: Grade 3 to 1 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 3 to 2 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 3 to 3 | 0 | 0 | 0
  Leukocytosis: Grade 3 to 4 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 4 to 0 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 4 to 1 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 4 to 2 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 4 to 3 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Leukocytosis: Grade 4 to 4 | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis. | NA — Grade 1 and Grade 2 are not defined in CTCAE (i.e. Blank) and Grade 4 only includes non-quantitative conditions, therefore Grades 1, 2 and 4 are NA for Leukocytosis.
  Lymphocyte count decreased: Grade 0 to 0 | 0 | 0 | 3
  Lymphocyte count decreased: Grade 0 to 1 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 0 to 2 | 0 | 0 | 2
  Lymphocyte count decreased: Grade 0 to 3 | 1 | 1 | 0
  Lymphocyte count decreased: Grade 0 to 4 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 1 to 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 1 to 1 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 1 to 2 | 0 | 1 | 0
  Lymphocyte count decreased: Grade 1 to 3 | 1 | 0 | 1
  Lymphocyte count decreased: Grade 1 to 4 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 2 to 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 2 to 1 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 2 to 2 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 2 to 3 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 2 to 4 | 1 | 0 | 0
  Lymphocyte count decreased: Grade 3 to 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 3 to 1 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 3 to 2 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 3 to 3 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 3 to 4 | 0 | 0 | 1
  Lymphocyte count decreased: Grade 4 to 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 4 to 1 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 4 to 2 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 4 to 3 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 4 to 4 | 0 | 0 | 0
  Lymphocyte count increased: Grade 0 to 0 | 3 | 2 | 7
  Lymphocyte count increased: Grade 0 to 1 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 0 to 2 | 0 | 0 | 0
  Lymphocyte count increased: Grade 0 to 3 | 0 | 0 | 0
  Lymphocyte count increased: Grade 0 to 4 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 1 to 0 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 1 to 1 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 1 to 2 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 1 to 3 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 1 to 4 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 2 to 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 2 to 1 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 2 to 2 | 0 | 0 | 0
  Lymphocyte count increased: Grade 2 to 3 | 0 | 0 | 0
  Lymphocyte count increased: Grade 2 to 4 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 3 to 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 3 to 1 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 3 to 2 | 0 | 0 | 0
  Lymphocyte count increased: Grade 3 to 3 | 0 | 0 | 0
  Lymphocyte count increased: Grade 3 to 4 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 4 to 0 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 4 to 1 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 4 to 2 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 4 to 3 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Lymphocyte count increased: Grade 4 to 4 | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased. | NA — Grade 1 and Grade 4 are not defined in CTCAE (i.e. Blank), therefore, Grades 1 and 4 are NA for lymphocyte count increased.
  Neutrophil count decrease: Grade 0 to 0 | 2 | 2 | 7
  Neutrophil count decrease: Grade 0 to 1 | 0 | 0 | 0
  Neutrophil count decrease: Grade 0 to 2 | 1 | 0 | 0
  Neutrophil count decrease: Grade 0 to 3 | 0 | 0 | 0
  Neutrophil count decrease: Grade 0 to 4 | 0 | 0 | 0
  Neutrophil count decrease: Grade 1 to 0 | 0 | 0 | 0
  Neutrophil count decrease: Grade 1 to 1 | 0 | 0 | 0
  Neutrophil count decrease: Grade 1 to 2 | 0 | 0 | 0
  Neutrophil count decrease: Grade 1 to 3 | 0 | 0 | 0
  Neutrophil count decrease: Grade 1 to 4 | 0 | 0 | 0
  Neutrophil count decrease: Grade 2 to 0 | 0 | 0 | 0
  Neutrophil count decrease: Grade 2 to 1 | 0 | 0 | 0
  Neutrophil count decrease: Grade 2 to 2 | 0 | 0 | 0
  Neutrophil count decrease: Grade 2 to 3 | 0 | 0 | 0
  Neutrophil count decrease: Grade 2 to 4 | 0 | 0 | 0
  Neutrophil count decrease: Grade 3 to 0 | 0 | 0 | 0
  Neutrophil count decrease: Grade 3 to 1 | 0 | 0 | 0
  Neutrophil count decrease: Grade 3 to 2 | 0 | 00 | 0
  Neutrophil count decrease: Grade 3 to 3 | 0 | 0 | 0
  Neutrophil count decrease: Grade 3 to 4 | 0 | 0 | 0
  Neutrophil count decrease: Grade 4 to 0 | 0 | 0 | 0
  Neutrophil count decrease: Grade 4 to 1 | 0 | 0 | 0
  Neutrophil count decrease: Grade 4 to 2 | 0 | 0 | 0
  Neutrophil count decrease: Grade 4 to 3 | 0 | 0 | 0
  Neutrophil count decrease: Grade 4 to 4 | 0 | 0 | 0
  Platelet count decreased: Grade 0 to 0 | 2 | 2 | 6
  Platelet count decreased: Grade 0 to 1 | 0 | 0 | 0
  Platelet count decreased: Grade 0 to 2 | 1 | 0 | 1
  Platelet count decreased: Grade 0 to 3 | 0 | 0 | 0
  Platelet count decreased: Grade 0 to 4 | 0 | 0 | 0
  Platelet count decreased: Grade 1 to 0 | 0 | 0 | 0
  Platelet count decreased: Grade 1 to 1 | 0 | 0 | 0
  Platelet count decreased: Grade 1 to 2 | 0 | 0 | 0
  Platelet count decreased: Grade 1 to 3 | 0 | 0 | 0
  Platelet count decreased: Grade 1 to 4 | 0 | 0 | 0
  Platelet count decreased: Grade 2 to 0 | 0 | 0 | 0
  Platelet count decreased: Grade 2 to 1 | 0 | 0 | 0
  Platelet count decreased: Grade 2 to 2 | 0 | 0 | 0
  Platelet count decreased: Grade 2 to 3 | 0 | 0 | 0
  Platelet count decreased: Grade 2 to 4 | 0 | 0 | 0
  Platelet count decreased: Grade 3 to 0 | 0 | 0 | 0
  Platelet count decreased: Grade 3 to 1 | 0 | 0 | 0
  Platelet count decreased: Grade 3 to 2 | 0 | 0 | 0
  Platelet count decreased: Grade 3 to 3 | 0 | 0 | 0
  Platelet count decreased: Grade 3 to 4 | 0 | 0 | 0
  Platelet count decreased: Grade 4 to 0 | 0 | 0 | 0
  Platelet count decreased: Grade 4 to 1 | 0 | 0 | 0
  Platelet count decreased: Grade 4 to 2 | 0 | 0 | 0
  Platelet count decreased: Grade 4 to 3 | 0 | 0 | 0
  Platelet count decreased: Grade 4 to 4 | 0 | 0 | 0
  White blood Cell decreased: Grade 0 to 0 | 1 | 1 | 5
  White blood Cell decreased: Grade 0 to 1 | 1 | 0 | 2
  White blood Cell decreased: Grade 0 to 2 | 0 | 0 | 0
  White blood Cell decreased: Grade 0 to 3 | 1 | 0 | 0
  White blood Cell decreased: Grade 0 to 4 | 0 | 0 | 0
  White blood Cell decreased: Grade 1 to 0 | 0 | 0 | 0
  White blood Cell decreased: Grade 1 to 1 | 0 | 1 | 0
  White blood Cell decreased: Grade 1 to 2 | 0 | 0 | 0
  White blood Cell decreased: Grade 1 to 3 | 0 | 0 | 0
  White blood Cell decreased: Grade 1 to 4 | 0 | 0 | 0
  White blood Cell decreased: Grade 2 to 0 | 0 | 0 | 0
  White blood Cell decreased: Grade 2 to 1 | 0 | 0 | 0
  White blood Cell decreased: Grade 2 to 2 | 0 | 0 | 0
  White blood Cell decreased: Grade 2 to 3 | 0 | 0 | 0
  White blood Cell decreased: Grade 2 to 4 | 0 | 0 | 0
  White blood Cell decreased: Grade 3 to 0 | 0 | 0 | 0
  White blood Cell decreased: Grade 3 to 1 | 0 | 0 | 0
  White blood Cell decreased: Grade 3 to 2 | 0 | 0 | 0
  White blood Cell decreased: Grade 3 to 3 | 0 | 0 | 0
  White blood Cell decreased: Grade 3 to 4 | 0 | 0 | 0
  White blood Cell decreased: Grade 4 to 0 | 0 | 0 | 0
  White blood Cell decreased: Grade 4 to 1 | 0 | 0 | 0
  White blood Cell decreased: Grade 4 to 2 | 0 | 0 | 0
  White blood Cell decreased: Grade 4 to 3 | 0 | 0 | 0
  White blood Cell decreased: Grade 4 to 4 | 0 | 0 | 0

39. Secondary Outcome: Phase 2 of Sub-Study B: Number of Participants With Shift From Baseline in Chemistry Parameter Values Based on CTCAE V5.0
Description: Chemistry parameters included: ALT increased, ALP increased, AST increased, blood bilirubin increased, chronic kidney disease, creatinine increased, hypercalcemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypokalemia, hypomagnesemia, hyponatremia, lipase increased, serum amylase increased. Number of participants with maximum CTCAE V5.0 grade in chemistry parameters were reported. Grade 0= non-missing lab value that does not meet either of Grade 1 through 4 criteria; Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling.
Time Frame: as for outcome 5
Population: Safety analysis set included all participants who received at least 1 dose of study drug. Here, "Number Analyzed" signifies number of participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
Number analyzed (Participants) | 3 | 2 | 7
Participants
  ALT increased: Grade 0 to 0 | 1 | 1 | 3
  ALT increased: Grade 0 to 1 | 1 | 0 | 3
  ALT increased: Grade 0 to 2 | 0 | 0 | 0
  ALT increased: Grade 0 to 3 | 1 | 1 | 0
  ALT increased: Grade 0 to 4 | 0 | 0 | 1
  ALT increased: Grade 1 to 0 | 0 | 0 | 0
  ALT increased: Grade 1 to 1 | 0 | 0 | 0
  ALT increased: Grade 1 to 2 | 0 | 0 | 0
  ALT increased: Grade 1 to 3 | 0 | 0 | 0
  ALT increased: Grade 1 to 4 | 0 | 0 | 0
  ALT increased: Grade 2 to 0 | 0 | 0 | 0
  ALT increased: Grade 2 to 1 | 0 | 0 | 0
  ALT increased: Grade 2 to 2 | 0 | 0 | 0
  ALT increased: Grade 2 to 3 | 0 | 0 | 0
  ALT increased: Grade 2 to 4 | 0 | 0 | 0
  ALT increased: Grade 3 to 0 | 0 | 0 | 0
  ALT increased: Grade 3 to 1 | 0 | 0 | 0
  ALT increased: Grade 3 to 2 | 0 | 0 | 0
  ALT increased: Grade 3 to 3 | 0 | 0 | 0
  ALT increased: Grade 3 to 4 | 0 | 0 | 0
  ALT increased: Grade 4 to 0 | 0 | 0 | 0
  ALT increased: Grade 4 to 1 | 0 | 0 | 0
  ALT increased: Grade 4 to 2 | 0 | 0 | 0
  ALT increased: Grade 4 to 3 | 0 | 0 | 0
  ALT increased: Grade 4 to 4 | 0 | 0 | 0
  ALP increased: Grade 0 to 0 | 0 | 1 | 3
  ALP increased: Grade 0 to 1 | 2 | 1 | 2
  ALP increased: Grade 0 to 2 | 0 | 0 | 0
  ALP increased: Grade 0 to 3 | 0 | 0 | 0
  ALP increased: Grade 0 to 4 | 0 | 0 | 0
  ALP increased: Grade 1 to 0 | 1 | 0 | 2
  ALP increased: Grade 1 to 1 | 0 | 0 | 0
  ALP increased: Grade 1 to 2 | 0 | 0 | 0
  ALP increased: Grade 1 to 3 | 0 | 0 | 0
  ALP increased: Grade 1 to 4 | 0 | 0 | 0
  ALP increased: Grade 2 to 0 | 0 | 0 | 0
  ALP increased: Grade 2 to 1 | 0 | 0 | 0
  ALP increased: Grade 2 to 2 | 0 | 0 | 0
  ALP increased: Grade 2 to 3 | 0 | 0 | 0
  ALP increased: Grade 2 to 4 | 0 | 0 | 0
  ALP increased: Grade 3 to 0 | 0 | 0 | 0
  ALP increased: Grade 3 to 1 | 0 | 0 | 0
  ALP increased: Grade 3 to 2 | 0 | 0 | 0
  ALP increased: Grade 3 to 3 | 0 | 0 | 0
  ALP increased: Grade 3 to 4 | 0 | 0 | 0
  ALP increased: Grade 4 to 0 | 0 | 0 | 0
  ALP increased: Grade 4 to 1 | 0 | 0 | 0
  ALP increased: Grade 4 to 2 | 0 | 0 | 0
  ALP increased: Grade 4 to 3 | 0 | 0 | 0
  ALP increased: Grade 4 to 4 | 0 | 0 | 0
  AST increase: Grade 0 to 0 | 1 | 1 | 2
  AST increase: Grade 0 to 1 | 1 | 0 | 4
  AST increase: Grade 0 to 2 | 0 | 0 | 0
  AST increase: Grade 0 to 3 | 1 | 1 | 0
  AST increase: Grade 0 to 4 | 0 | 0 | 1
  AST increase: Grade 1 to 0 | 0 | 0 | 0
  AST increase: Grade 1 to 1 | 0 | 0 | 0
  AST increase: Grade 1 to 2 | 0 | 0 | 0
  AST increase: Grade 1 to 3 | 0 | 0 | 0
  AST increase: Grade 1 to 4 | 0 | 0 | 0
  AST increase: Grade 2 to 0 | 0 | 0 | 0
  AST increase: Grade 2 to 1 | 0 | 0 | 0
  AST increase: Grade 2 to 2 | 0 | 0 | 0
  AST increase: Grade 2 to 3 | 0 | 0 | 0
  AST increase: Grade 2 to 4 | 0 | 0 | 0
  AST increase: Grade 3 to 0 | 0 | 0 | 0
  AST increase: Grade 3 to 1 | 0 | 0 | 0
  AST increase: Grade 3 to 2 | 0 | 0 | 0
  AST increase: Grade 3 to 3 | 0 | 0 | 0
  AST increase: Grade 3 to 4 | 0 | 0 | 0
  AST increase: Grade 4 to 0 | 0 | 0 | 0
  AST increase: Grade 4 to 1 | 0 | 0 | 0
  AST increase: Grade 4 to 2 | 0 | 0 | 0
  AST increase: Grade 4 to 3 | 0 | 0 | 0
  AST increase: Grade 4 to 4 | 0 | 0 | 0
  Blood bilirubin increased: Grade 0 to 0 | 2 | 1 | 6
  Blood bilirubin increased: Grade 0 to 1 | 1 | 1 | 0
  Blood bilirubin increased: Grade 0 to 2 | 0 | 0 | 0
  Blood bilirubin increased: Grade 0 to 3 | 0 | 0 | 1
  Blood bilirubin increased: Grade 0 to 4 | 0 | 0 | 0
  Blood bilirubin increased: Grade 1 to 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 1 to 1 | 0 | 0 | 0
  Blood bilirubin increased: Grade 1 to 2 | 0 | 0 | 0
  Blood bilirubin increased: Grade 1 to 3 | 0 | 0 | 0
  Blood bilirubin increased: Grade 1 to 4 | 0 | 0 | 0
  Blood bilirubin increased: Grade 2 to 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 2 to 1 | 0 | 0 | 0
  Blood bilirubin increased: Grade 2 to 2 | 0 | 0 | 0
  Blood bilirubin increased: Grade 2 to 3 | 0 | 0 | 0
  Blood bilirubin increased: Grade 2 to 4 | 0 | 0 | 0
  Blood bilirubin increased: Grade 3 to 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 3 to 1 | 0 | 0 | 0
  Blood bilirubin increased: Grade 3 to 2 | 0 | 0 | 0
  Blood bilirubin increased: Grade 3 to 3 | 0 | 0 | 0
  Blood bilirubin increased: Grade 3 to 4 | 0 | 0 | 0
  Blood bilirubin increased: Grade 4 to 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 4 to 1 | 0 | 0 | 0
  Blood bilirubin increased: Grade 4 to 2 | 0 | 0 | 0
  Blood bilirubin increased: Grade 4 to 3 | 0 | 0 | 0
  Blood bilirubin increased: Grade 4 to 4 | 0 | 0 | 0
  CPK increased: number analyzed (Participants) | 3 | 2 | 6
  CPK increased: Grade 0 to 0 | 3 | 2 | 5
  CPK increased: Grade 0 to 1 | 0 | 0 | 0
  CPK increased: Grade 0 to 2 | 0 | 0 | 0
  CPK increased: Grade 0 to 3 | 0 | 0 | 0
  CPK increased: Grade 0 to 4 | 0 | 0 | 0
  CPK increased: Grade 1 to 0 | 0 | 0 | 1
  CPK increased: Grade 1 to 1 | 0 | 0 | 0
  CPK increased: Grade 1 to 2 | 0 | 0 | 0
  CPK increased: Grade 1 to 3 | 0 | 0 | 0
  CPK increased: Grade 1 to 4 | 0 | 0 | 0
  CPK increased: Grade 2 to 0 | 0 | 0 | 0
  CPK increased: Grade 2 to 1 | 0 | 0 | 0
  CPK increased: Grade 2 to 2 | 0 | 0 | 0
  CPK increased: Grade 2 to 3 | 0 | 0 | 0
  CPK increased: Grade 2 to 4 | 0 | 0 | 0
  CPK increased: Grade 3 to 0 | 0 | 0 | 0
  CPK increased: Grade 3 to 1 | 0 | 0 | 0
  CPK increased: Grade 3 to 2 | 0 | 0 | 0
  CPK increased: Grade 3 to 3 | 0 | 0 | 0
  CPK increased: Grade 3 to 4 | 0 | 0 | 0
  CPK increased: Grade 4 to 0 | 0 | 0 | 0
  CPK increased: Grade 4 to 1 | 0 | 0 | 0
  CPK increased: Grade 4 to 2 | 0 | 0 | 0
  CPK increased: Grade 4 to 3 | 0 | 0 | 0
  CPK increased: Grade 4 to 4 | 0 | 0 | 0
  Chronic kidney disease: Grade 0 to 0 | 1 | 2 | 5
  Chronic kidney disease: Grade 0 to 1 | 0 | 0 | 0
  Chronic kidney disease: Grade 0 to 2 | 0 | 0 | 1
  Chronic kidney disease: Grade 0 to 3 | 1 | 0 | 0
  Chronic kidney disease: Grade 0 to 4 | 0 | 0 | 0
  Chronic kidney disease: Grade 1 to 0 | 0 | 0 | 0
  Chronic kidney disease: Grade 1 to 1 | 0 | 0 | 0
  Chronic kidney disease: Grade 1 to 2 | 1 | 0 | 0
  Chronic kidney disease: Grade 1 to 3 | 0 | 0 | 0
  Chronic kidney disease: Grade 1 to 4 | 0 | 0 | 0
  Chronic kidney disease: Grade 2 to 0 | 0 | 0 | 0
  Chronic kidney disease: Grade 2 to 1 | 0 | 0 | 0
  Chronic kidney disease: Grade 2 to 2 | 0 | 0 | 1
  Chronic kidney disease: Grade 2 to 3 | 0 | 0 | 0
  Chronic kidney disease: Grade 2 to 4 | 0 | 0 | 0
  Chronic kidney disease: Grade 3 to 0 | 0 | 0 | 0
  Chronic kidney disease: Grade 3 to 1 | 0 | 0 | 0
  Chronic kidney disease: Grade 3 to 2 | 0 | 0 | 0
  Chronic kidney disease: Grade 3 to 3 | 0 | 0 | 0
  Chronic kidney disease: Grade 3 to 4 | 0 | 0 | 0
  Chronic kidney disease: Grade 4 to 0 | 0 | 0 | 0
  Chronic kidney disease: Grade 4 to 1 | 0 | 0 | 0
  Chronic kidney disease: Grade 4 to 2 | 0 | 0 | 0
  Chronic kidney disease: Grade 4 to 3 | 0 | 0 | 0
  Chronic kidney disease: Grade 4 to 4 | 0 | 00 | 0
  Creatinine increased: Grade 0 to 0 | 1 | 2 | 5
  Creatinine increased: Grade 0 to 1 | 0 | 0 | 1
  Creatinine increased: Grade 0 to 2 | 0 | 0 | 0
  Creatinine increased: Grade 0 to 3 | 1 | 0 | 0
  Creatinine increased: Grade 0 to 4 | 0 | 0 | 0
  Creatinine increased: Grade 1 to 0 | 0 | 0 | 0
  Creatinine increased: Grade 1 to 1 | 1 | 0 | 1
  Creatinine increased: Grade 1 to 2 | 0 | 0 | 0
  Creatinine increased: Grade 1 to 3 | 0 | 0 | 0
  Creatinine increased: Grade 1 to 4 | 0 | 0 | 0
  Creatinine increased: Grade 2 to 0 | 0 | 0 | 0
  Creatinine increased: Grade 2 to 1 | 0 | 0 | 0
  Creatinine increased: Grade 2 to 2 | 0 | 0 | 0
  Creatinine increased: Grade 2 to 3 | 0 | 0 | 0
  Creatinine increased: Grade 2 to 4 | 0 | 0 | 0
  Creatinine increased: Grade 3 to 0 | 0 | 0 | 0
  Creatinine increased: Grade 3 to 1 | 0 | 0 | 0
  Creatinine increased: Grade 3 to 2 | 0 | 0 | 0
  Creatinine increased: Grade 3 to 3 | 0 | 0 | 0
  Creatinine increased: Grade 3 to 4 | 0 | 0 | 0
  Creatinine increased: Grade 4 to 0 | 0 | 0 | 0
  Creatinine increased: Grade 4 to 1 | 0 | 0 | 0
  Creatinine increased: Grade 4 to 2 | 0 | 0 | 0
  Creatinine increased: Grade 4 to 3 | 0 | 0 | 0
  Creatinine increased: Grade 4 to 4 | 0 | 0 | 0
  Hypercalcemia: Grade 0 to 0 | 2 | 2 | 7
  Hypercalcemia: Grade 0 to 1 | 1 | 0 | 0
  Hypercalcemia: Grade 0 to 2 | 0 | 0 | 0
  Hypercalcemia: Grade 0 to 3 | 0 | 0 | 0
  Hypercalcemia: Grade 0 to 4 | 0 | 0 | 0
  Hypercalcemia: Grade 1 to 0 | 0 | 0 | 0
  Hypercalcemia: Grade 1 to 1 | 0 | 0 | 0
  Hypercalcemia: Grade 1 to 2 | 0 | 0 | 0
  Hypercalcemia: Grade 1 to 3 | 0 | 0 | 0
  Hypercalcemia: Grade 1 to 4 | 0 | 0 | 0
  Hypercalcemia: Grade 2 to 0 | 0 | 0 | 0
  Hypercalcemia: Grade 2 to 1 | 0 | 0 | 0
  Hypercalcemia: Grade 2 to 2 | 0 | 0 | 0
  Hypercalcemia: Grade 2 to 3 | 0 | 0 | 0
  Hypercalcemia: Grade 2 to 4 | 0 | 0 | 0
  Hypercalcemia: Grade 3 to 0 | 0 | 0 | 0
  Hypercalcemia: Grade 3 to 1 | 0 | 0 | 0
  Hypercalcemia: Grade 3 to 2 | 0 | 0 | 0
  Hypercalcemia: Grade 3 to 3 | 0 | 0 | 0
  Hypercalcemia: Grade 3 to 4 | 0 | 0 | 0
  Hypercalcemia: Grade 4 to 0 | 0 | 0 | 0
  Hypercalcemia: Grade 4 to 1 | 0 | 0 | 0
  Hypercalcemia: Grade 4 to 2 | 0 | 0 | 0
  Hypercalcemia: Grade 4 to 3 | 0 | 0 | 00
  Hypercalcemia: Grade 4 to 4 | 0 | 0 | 0
  Hyperkalemia: Grade 0 to 0 | 2 | 1 | 6
  Hyperkalemia: Grade 0 to 1 | 0 | 1 | 1
  Hyperkalemia: Grade 0 to 2 | 1 | 0 | 0
  Hyperkalemia: Grade 0 to 3 | 0 | 0 | 0
  Hyperkalemia: Grade 0 to 4 | 0 | 0 | 0
  Hyperkalemia: Grade 1 to 0 | 0 | 0 | 0
  Hyperkalemia: Grade 1 to 1 | 0 | 0 | 0
  Hyperkalemia: Grade 1 to 2 | 0 | 0 | 0
  Hyperkalemia: Grade 1 to 3 | 0 | 0 | 0
  Hyperkalemia: Grade 1 to 4 | 0 | 0 | 0
  Hyperkalemia: Grade 2 to 0 | 0 | 0 | 0
  Hyperkalemia: Grade 2 to 1 | 0 | 0 | 0
  Hyperkalemia: Grade 2 to 2 | 0 | 0 | 0
  Hyperkalemia: Grade 2 to 3 | 0 | 0 | 0
  Hyperkalemia: Grade 2 to 4 | 0 | 0 | 0
  Hyperkalemia: Grade 3 to 0 | 0 | 0 | 0
  Hyperkalemia: Grade 3 to 1 | 0 | 0 | 0
  Hyperkalemia: Grade 3 to 2 | 0 | 0 | 0
  Hyperkalemia: Grade 3 to 3 | 0 | 0 | 0
  Hyperkalemia: Grade 3 to 4 | 0 | 0 | 0
  Hyperkalemia: Grade 4 to 0 | 0 | 0 | 0
  Hyperkalemia: Grade 4 to 1 | 0 | 0 | 0
  Hyperkalemia: Grade 4 to 2 | 0 | 0 | 0
  Hyperkalemia: Grade 4 to 3 | 0 | 0 | 0
  Hyperkalemia: Grade 4 to 4 | 0 | 0 | 0
  Hypermagnesemia: Grade 0 to 0 | 3 | 2 | 6
  Hypermagnesemia: Grade 0 to 1 | 0 | 0 | 1
  Hypermagnesemia: Grade 0 to 2 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 0 to 3 | 0 | 0 | 0
  Hypermagnesemia: Grade 0 to 4 | 0 | 0 | 0
  Hypermagnesemia: Grade 1 to 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 1 to 1 | 0 | 0 | 0
  Hypermagnesemia: Grade 1 to 2 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 1 to 3 | 0 | 0 | 0
  Hypermagnesemia: Grade 1 to 4 | 0 | 0 | 0
  Hypermagnesemia: Grade 2 to 0 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 2 to 1 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 2 to 2 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 2 to 3 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 2 to 4 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 3 to 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 3 to 1 | 0 | 0 | 0
  Hypermagnesemia: Grade 3 to 2 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 3 to 3 | 0 | 0 | 0
  Hypermagnesemia: Grade 3 to 4 | 0 | 0 | 0
  Hypermagnesemia: Grade 4 to 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 4 to 1 | 0 | 0 | 0
  Hypermagnesemia: Grade 4 to 2 | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia. | NA — Grade 2 is not defined in CTCAE (i.e. Blank) therefore Grade 2 is NA for hypermagnesemia.
  Hypermagnesemia: Grade 4 to 3 | 0 | 0 | 0
  Hypermagnesemia: Grade 4 to 4 | 0 | 0 | 0
  Hypernatremia: Grade 0 to 0 | 3 | 2 | 6
  Hypernatremia: Grade 0 to 1 | 0 | 0 | 1
  Hypernatremia: Grade 0 to 2 | 0 | 0 | 0
  Hypernatremia: Grade 0 to 3 | 0 | 0 | 0
  Hypernatremia: Grade 0 to 4 | 0 | 0 | 0
  Hypernatremia: Grade 1 to 0 | 0 | 0 | 0
  Hypernatremia: Grade 1 to 1 | 0 | 0 | 0
  Hypernatremia: Grade 1 to 2 | 0 | 0 | 0
  Hypernatremia: Grade 1 to 3 | 0 | 0 | 0
  Hypernatremia: Grade 1 to 4 | 0 | 0 | 0
  Hypernatremia: Grade 2 to 0 | 0 | 0 | 0
  Hypernatremia: Grade 2 to 1 | 0 | 0 | 0
  Hypernatremia: Grade 2 to 2 | 0 | 0 | 0
  Hypernatremia: Grade 2 to 3 | 0 | 0 | 0
  Hypernatremia: Grade 2 to 4 | 0 | 0 | 0
  Hypernatremia: Grade 3 to 0 | 0 | 0 | 0
  Hypernatremia: Grade 3 to 1 | 0 | 0 | 0
  Hypernatremia: Grade 3 to 2 | 0 | 0 | 0
  Hypernatremia: Grade 3 to 3 | 0 | 0 | 0
  Hypernatremia: Grade 3 to 4 | 0 | 0 | 0
  Hypernatremia: Grade 4 to 0 | 0 | 0 | 0
  Hypernatremia: Grade 4 to 1 | 0 | 0 | 0
  Hypernatremia: Grade 4 to 2 | 0 | 0 | 0
  Hypernatremia: Grade 4 to 3 | 0 | 0 | 0
  Hypernatremia: Grade 4 to 4 | 0 | 0 | 0
  Hypoalbuminemia: Grade 0 to 0 | 1 | 2 | 4
  Hypoalbuminemia: Grade 0 to 1 | 1 | 0 | 1
  Hypoalbuminemia: Grade 0 to 2 | 1 | 0 | 2
  Hypoalbuminemia: Grade 0 to 3 | 0 | 0 | 0
  Hypoalbuminemia: Grade 0 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 1 to 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 1 to 1 | 0 | 0 | 0
  Hypoalbuminemia: Grade 1 to 2 | 0 | 0 | 0
  Hypoalbuminemia: Grade 1 to 3 | 0 | 0 | 0
  Hypoalbuminemia: Grade 1 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 2 to 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 2 to 1 | 0 | 0 | 0
  Hypoalbuminemia: Grade 2 to 2 | 0 | 0 | 0
  Hypoalbuminemia: Grade 2 to 3 | 0 | 0 | 0
  Hypoalbuminemia: Grade 2 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 3 to 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 3 to 1 | 0 | 0 | 0
  Hypoalbuminemia: Grade 3 to 2 | 0 | 0 | 0
  Hypoalbuminemia: Grade 3 to 3 | 0 | 0 | 0
  Hypoalbuminemia: Grade 3 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 4 to 0 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 4 to 1 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 4 to 2 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 4 to 3 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypoalbuminemia: Grade 4 to 4 | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia. | NA — Grade 4 only includes non-quantitative conditions; therefore Grade 4 is NA for hypoalbuminemia.
  Hypocalcemia: Grade 0 to 0 | 2 | 2 | 6
  Hypocalcemia: Grade 0 to 1 | 1 | 0 | 0
  Hypocalcemia: Grade 0 to 2 | 0 | 0 | 0
  Hypocalcemia: Grade 0 to 3 | 0 | 0 | 0
  Hypocalcemia: Grade 0 to 4 | 0 | 0 | 0
  Hypocalcemia: Grade 1 to 0 | 0 | 0 | 0
  Hypocalcemia: Grade 1 to 1 | 0 | 0 | 1
  Hypocalcemia: Grade 1 to 2 | 0 | 0 | 0
  Hypocalcemia: Grade 1 to 3 | 0 | 0 | 0
  Hypocalcemia: Grade 1 to 4 | 0 | 0 | 0
  Hypocalcemia: Grade 2 to 0 | 0 | 0 | 0
  Hypocalcemia: Grade 2 to 1 | 0 | 0 | 0
  Hypocalcemia: Grade 2 to 2 | 0 | 0 | 0
  Hypocalcemia: Grade 2 to 3 | 0 | 0 | 0
  Hypocalcemia: Grade 2 to 4 | 0 | 0 | 0
  Hypocalcemia: Grade 3 to 0 | 0 | 0 | 0
  Hypocalcemia: Grade 3 to 1 | 0 | 0 | 0
  Hypocalcemia: Grade 3 to 2 | 0 | 0 | 0
  Hypocalcemia: Grade 3 to 3 | 0 | 0 | 0
  Hypocalcemia: Grade 3 to 4 | 0 | 0 | 0
  Hypocalcemia: Grade 4 to 0 | 0 | 0 | 0
  Hypocalcemia: Grade 4 to 1 | 0 | 0 | 0
  Hypocalcemia: Grade 4 to 2 | 0 | 0 | 0
  Hypocalcemia: Grade 4 to 3 | 0 | 0 | 0
  Hypocalcemia: Grade 4 to 4 | 0 | 0 | 0
  Hypoglycemia: Grade 0 to 0 | 3 | 2 | 7
  Hypoglycemia: Grade 0 to 1 | 0 | 0 | 0
  Hypoglycemia: Grade 0 to 2 | 0 | 0 | 0
  Hypoglycemia: Grade 0 to 3 | 0 | 0 | 0
  Hypoglycemia: Grade 0 to 4 | 0 | 0 | 0
  Hypoglycemia: Grade 1 to 0 | 0 | 0 | 0
  Hypoglycemia: Grade 1 to 1 | 0 | 0 | 0
  Hypoglycemia: Grade 1 to 2 | 0 | 0 | 0
  Hypoglycemia: Grade 1 to 3 | 0 | 0 | 0
  Hypoglycemia: Grade 1 to 4 | 0 | 0 | 0
  Hypoglycemia: Grade 2 to 0 | 0 | 0 | 0
  Hypoglycemia: Grade 2 to 1 | 0 | 0 | 0
  Hypoglycemia: Grade 2 to 2 | 0 | 0 | 0
  Hypoglycemia: Grade 2 to 3 | 0 | 0 | 0
  Hypoglycemia: Grade 2 to 4 | 0 | 0 | 0
  Hypoglycemia: Grade 3 to 0 | 0 | 0 | 0
  Hypoglycemia: Grade 3 to 1 | 0 | 0 | 0
  Hypoglycemia: Grade 3 to 2 | 0 | 0 | 0
  Hypoglycemia: Grade 3 to 3 | 0 | 0 | 0
  Hypoglycemia: Grade 3 to 4 | 0 | 0 | 0
  Hypoglycemia: Grade 4 to 0 | 0 | 0 | 0
  Hypoglycemia: Grade 4 to 1 | 0 | 0 | 0
  Hypoglycemia: Grade 4 to 2 | 0 | 0 | 0
  Hypoglycemia: Grade 4 to 3 | 0 | 0 | 0
  Hypoglycemia: Grade 4 to 4 | 0 | 0 | 0
  Hypokalemia: Grade 0 to 0 | 2 | 1 | 4
  Hypokalemia: Grade 0 to 1 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 0 to 2 | 0 | 1 | 2
  Hypokalemia: Grade 0 to 3 | 1 | 0 | 0
  Hypokalemia: Grade 0 to 4 | 0 | 0 | 0
  Hypokalemia: Grade 1 to 0 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 1 to 1 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 1 to 2 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 1 to 3 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 1 to 4 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 2 to 0 | 0 | 0 | 0
  Hypokalemia: Grade 2 to 1 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 2 to 2 | 0 | 0 | 1
  Hypokalemia: Grade 2 to 3 | 0 | 0 | 0
  Hypokalemia: Grade 2 to 4 | 0 | 0 | 0
  Hypokalemia: Grade 3 to 0 | 0 | 0 | 0
  Hypokalemia: Grade 3 to 1 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 3 to 2 | 0 | 0 | 0
  Hypokalemia: Grade 3 to 3 | 0 | 0 | 0
  Hypokalemia: Grade 3 to 4 | 0 | 0 | 0
  Hypokalemia: Grade 4 to 0 | 0 | 0 | 0
  Hypokalemia: Grade 4 to 1 | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia. | NA — Grade 1 and Grade 2 are only distinguishable by non-quantitative conditions therefore Grade 1 is NA and values that could meet Grade 1 or Grade 2 criteria are presented as Grade 2 for hypokalemia.
  Hypokalemia: Grade 4 to 2 | 0 | 0 | 0
  Hypokalemia: Grade 4 to 3 | 0 | 0 | 0
  Hypokalemia: Grade 4 to 4 | 0 | 0 | 0
  Hypomagnesemia: Grade 0 to 0 | 2 | 2 | 3
  Hypomagnesemia: Grade 0 to 1 | 0 | 0 | 4
  Hypomagnesemia: Grade 0 to 2 | 1 | 0 | 0
  Hypomagnesemia: Grade 0 to 3 | 0 | 0 | 0
  Hypomagnesemia: Grade 0 to 4 | 0 | 0 | 0
  Hypomagnesemia: Grade 1 to 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 1 to 1 | 0 | 0 | 0
  Hypomagnesemia: Grade 1 to 2 | 0 | 0 | 0
  Hypomagnesemia: Grade 1 to 3 | 0 | 0 | 0
  Hypomagnesemia: Grade 1 to 4 | 0 | 0 | 0
  Hypomagnesemia: Grade 2 to 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 2 to 1 | 0 | 0 | 0
  Hypomagnesemia: Grade 2 to 2 | 0 | 0 | 0
  Hypomagnesemia: Grade 2 to 3 | 0 | 0 | 0
  Hypomagnesemia: Grade 2 to 4 | 0 | 0 | 0
  Hypomagnesemia: Grade 3 to 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 3 to 1 | 0 | 0 | 0
  Hypomagnesemia: Grade 3 to 2 | 0 | 0 | 0
  Hypomagnesemia: Grade 3 to 3 | 0 | 0 | 0
  Hypomagnesemia: Grade 3 to 4 | 0 | 0 | 0
  Hypomagnesemia: Grade 4 to 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 4 to 1 | 0 | 0 | 0
  Hypomagnesemia: Grade 4 to 2 | 0 | 0 | 0
  Hypomagnesemia: Grade 4 to 3 | 0 | 0 | 0
  Hypomagnesemia: Grade 4 to 4 | 0 | 0 | 0
  Hyponatremia: Grade 0 to 0 | 2 | 1 | 4
  Hyponatremia: Grade 0 to 1 | 1 | 0 | 0
  Hyponatremia: Grade 0 to 2 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 0 to 3 | 0 | 0 | 3
  Hyponatremia: Grade 0 to 4 | 0 | 0 | 0
  Hyponatremia: Grade 1 to 0 | 0 | 0 | 0
  Hyponatremia: Grade 1 to 1 | 0 | 0 | 0
  Hyponatremia: Grade 1 to 2 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 1 to 3 | 0 | 1 | 0
  Hyponatremia: Grade 1 to 4 | 0 | 0 | 0
  Hyponatremia: Grade 2 to 0 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 2 to 1 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 2 to 2 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 2 to 3 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 2 to 4 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 3 to 0 | 0 | 0 | 0
  Hyponatremia: Grade 3 to 1 | 0 | 0 | 0
  Hyponatremia: Grade 3 to 2 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 3 to 3 | 0 | 0 | 0
  Hyponatremia: Grade 3 to 4 | 0 | 0 | 0
  Hyponatremia: Grade 4 to 0 | 0 | 0 | 0
  Hyponatremia: Grade 4 to 1 | 0 | 0 | 0
  Hyponatremia: Grade 4 to 2 | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia. | NA — Grade 2 and Grade 3 are only distinguishable by non-quantitative conditions therefore Grade 2 is NA and values that could meet Grade 2 or Grade 3 criteria are presented as Grade 3 for hyponatremia.
  Hyponatremia: Grade 4 to 3 | 0 | 0 | 0
  Hyponatremia: Grade 4 to 4 | 0 | 0 | 0
  Lipase increased: Grade 0 to 0 | 1 | 2 | 5
  Lipase increased: Grade 0 to 1 | 2 | 0 | 0
  Lipase increased: Grade 0 to 2 | 0 | 0 | 1
  Lipase increased: Grade 0 to 3 | 0 | 0 | 1
  Lipase increased: Grade 0 to 4 | 0 | 0 | 0
  Lipase increased: Grade 1 to 0 | 0 | 0 | 0
  Lipase increased: Grade 1 to 1 | 0 | 0 | 0
  Lipase increased: Grade 1 to 2 | 0 | 0 | 0
  Lipase increased: Grade 1 to 3 | 0 | 0 | 0
  Lipase increased: Grade 1 to 4 | 0 | 0 | 0
  Lipase increased: Grade 2 to 0 | 0 | 0 | 0
  Lipase increased: Grade 2 to 1 | 0 | 0 | 0
  Lipase increased: Grade 2 to 2 | 0 | 0 | 0
  Lipase increased: Grade 2 to 3 | 0 | 0 | 0
  Lipase increased: Grade 2 to 4 | 0 | 0 | 0
  Lipase increased: Grade 3 to 0 | 0 | 0 | 0
  Lipase increased: Grade 3 to 1 | 0 | 0 | 0
  Lipase increased: Grade 3 to 2 | 0 | 0 | 0
  Lipase increased: Grade 3 to 3 | 0 | 0 | 0
  Lipase increased: Grade 3 to 4 | 0 | 0 | 0
  Lipase increased: Grade 4 to 0 | 0 | 0 | 0
  Lipase increased: Grade 4 to 1 | 0 | 0 | 0
  Lipase increased: Grade 4 to 2 | 0 | 0 | 0
  Lipase increased: Grade 4 to 3 | 0 | 0 | 0
  Lipase increased: Grade 4 to 4 | 0 | 0 | 0
  Serum amylase increased: Grade 0 to 0 | 2 | 2 | 4
  Serum amylase increased: Grade 0 to 1 | 1 | 0 | 1
  Serum amylase increased: Grade 0 to 2 | 0 | 0 | 0
  Serum amylase increased: Grade 0 to 3 | 0 | 0 | 0
  Serum amylase increased: Grade 0 to 4 | 0 | 0 | 0
  Serum amylase increased: Grade 1 to 0 | 0 | 0 | 0
  Serum amylase increased: Grade 1 to 1 | 0 | 0 | 0
  Serum amylase increased: Grade 1 to 2 | 0 | 0 | 0
  Serum amylase increased: Grade 1 to 3 | 0 | 0 | 0
  Serum amylase increased: Grade 1 to 4 | 0 | 0 | 0
  Serum amylase increased: Grade 2 to 0 | 0 | 0 | 0
  Serum amylase increased: Grade 2 to 1 | 0 | 0 | 0
  Serum amylase increased: Grade 2 to 2 | 0 | 0 | 1
  Serum amylase increased: Grade 2 to 3 | 0 | 0 | 1
  Serum amylase increased: Grade 2 to 4 | 0 | 0 | 0
  Serum amylase increased: Grade 3 to 0 | 0 | 0 | 0
  Serum amylase increased: Grade 3 to 1 | 0 | 0 | 0
  Serum amylase increased: Grade 3 to 2 | 0 | 0 | 0
  Serum amylase increased: Grade 3 to 3 | 0 | 0 | 0
  Serum amylase increased: Grade 3 to 4 | 0 | 0 | 0
  Serum amylase increased: Grade 4 to 0 | 0 | 0 | 0
  Serum amylase increased: Grade 4 to 1 | 0 | 0 | 0
  Serum amylase increased: Grade 4 to 2 | 0 | 0 | 0
  Serum amylase increased: Grade 4 to 3 | 0 | 0 | 0
  Serum amylase increased: Grade 4 to 4 | 0 | 0 | 0

40. Secondary Outcome: Phase 1b of Sub-Study B: Objective Response Rate
Description: ORR was defined as percentage of participants with confirmed CR or PR according to RECIST v1.1 based on investigator assessment, from the date of first CR or PR until the date of the first documentation of PD, death, or start of new anticancer therapy. CR was defined as complete disappearance of all target lesions with exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. PD was defined as 20% increase in sum of diameters of target measurable lesions above smallest sum observed (over baseline if no decrease in the sum was observed during therapy), with a minimum absolute increase of 5 mm. Two sided 95% CI was based on Clopper-Pearson method.
Time Frame: From the date of first CR or PR until the date of the first documentation of PD, death, or start of new anticancer therapy, whichever occurred first (maximum of 21 months)
Population: Full analysis set included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg)
Number analyzed (Participants) | 3 | 6
Percentage of participants | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 45.9]

41. Secondary Outcome: Phase 1b of Sub-Study B: Duration of Response (DR)
Description: DR was defined for participants with confirmed objective response (OR) as time from date of first documentation of OR to the date of first documentation of PD or death (any cause), whichever occurred first. OR=CR or PR according to RECIST v1.1 based on investigator assessment. CR and PR must be confirmed by repeat assessments performed no <4 weeks after criteria for response were first met. CR=complete disappearance of all target lesions (TLs) with exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). PR=greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions (TMLs). PD=20% increase in sum of diameters of TMLs above smallest sum observed (over baseline if no decrease in sum was observed during therapy), with a minimum absolute increase of 5 mm.
Time Frame: From the date of first documentation of OR to the date of first documentation of PD or death, whichever occurred first (maximum of 21 months)
Population: Data was not estimable due to insufficient number of participants (with events) evaluable for this outcome measure.
Arm/Group | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg)
Number analyzed (Participants) | 0 | 0

42. Secondary Outcome: Phase 1b of Sub-Study B: Time to Tumor Response (TTR)
Description: as for outcome 14
Time Frame: From the date of first dose of study treatment to the date of first documentation of objective response (CR or PR) (maximum of 21 months)
Population: Data was not estimable due to insufficient number of participants (with events) evaluable for this outcome measure.
Arm/Group | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg)
Number analyzed (Participants) | 0 | 0

43. Secondary Outcome: Phase 1b of Sub-Study B: Progression-Free Survival (PFS)
Description: as for outcome 15
Time Frame: From the date of first dose of study treatment to the date of first documentation of PD or death due to any cause, whichever occurred first (maximum of 21 months)
Population: Full analysis set included all participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg)
Number analyzed (Participants) | 3 | 6
Months | 3.6 [0.7 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with event. | 6.5 [3.6 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with event.

44. Secondary Outcome: Phase 2 of Sub-Study B: Duration of Response (DR)
Description: as for outcome 13
Time Frame: From date of first documentation of OR to the date of first documentation of PD or death, whichever occurred first (maximum of 21 months)
Population: Full analysis set included all participants who received at least 1 dose of study drug. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and included only those participants with confirmed OR.'
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
Number analyzed (Participants) | 1 | 1 | 1
Months | NA [NA to NA] — Median and 95% CI could not be calculated as the only participant analyzed did not have an event of interest. | NA [NA to NA] — Median and 95% CI could not be calculated as the only participant analyzed did not have an event of interest. | 5.8 [NA to NA] — 95% CI could not be calculated because there was only one patient analyzed.

45. Secondary Outcome: Phase 2 of Sub-Study B: Time to Tumor Response (TTR)
Description: TTR is defined for participants with confirmed OR as the time from the date of first dose of study treatment to the date of first documentation of objective response (CR or PR) which was subsequently confirmed. CR=complete disappearance of all target lesions with exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). PR=greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions.
Time Frame: as for outcome 42
Population: Full analysis set included all participants who received at least 1 dose of study drug. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
Number analyzed (Participants) | 1 | 1 | 1
Months | 4.1 [4.1 to 4.1] | 1.3 [1.3 to 1.3] | 1.4 [1.4 to 1.4]

46. Secondary Outcome: Phase 2 of Sub-Study B: Progression-Free Survival (PFS)
Description: as for outcome 15
Time Frame: as for outcome 43
Population: Full analysis set included all participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
Number analyzed (Participants) | 3 | 2 | 7
Months | 4.2 [4.0 to NA] — Upper limit of 95% CI could not be calculated due to insufficient participants with event. | NA [2.8 to NA] — Median and upper limit of 95% CI could not be calculated due to insufficient participants with event. | 3.4 [1.4 to NA] — Upper limit of 95% CI could not be calculated due to insufficient participants with event.

47. Secondary Outcome: Phase 2 of Sub-Study B: Overall Survival (OS)
Description: as for outcome 16
Time Frame: From the date of first dose of study treatment to the date of death due to any cause or censoring date, whichever occurred first (maximum of 21 months)
Population: Full analysis set included all participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
Number analyzed (Participants) | 3 | 2 | 7
Months | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient participants with event. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient participants with event. | 4.0 [NA to NA] — Upper and lower limits of 95% CI could not be calculated due to insufficient participants with event.

48. Secondary Outcome: Phase 1b of Sub-Study B: Cmax of Sasanlimab
Time Frame: Cycle 1: pre-dose, 168 hours post-dose on Day 1, Cycle 5: pre-dose, 168 hours post-dose on Day 1 (1 cycle= 21 days)
Population: PK parameter analysis set was subset of safety analysis set (participants who received at least 1 dose of study drug) with participants who had at least 1 of PK parameters of interest for measured analytes related to study drug (i.e., sasanlimab). Here, ''Number of Participants Analyzed'' signifies participants evaluable for this outcome measure. Here, 'Number Analyzed' signifies participants evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg)
Number analyzed (Participants) | 3 | 3
Nanograms per milliliter
  Cycle 1 | 8840 (127) | 11570 (79)
  Cycle 5: number analyzed (Participants) | 2 | 3
  Cycle 5 | 23080 (NA) — Geometric coefficient of variation could not be calculated as at least 3 values were required and this criterion could not be fulfilled due to lack of available data. | 47340 (42)

49. Secondary Outcome: Phase 1b of Sub-Study B: Cmax of Axitinib
Time Frame: Cycle 1: pre-dose on Day 1, Day 8 and 3 hours post-dose on Day 1; Cycle 5: pre-dose on Day 1, Day 8 and 3 hours post-dose on Day 1 (1 cycle= 21 days)
Population: PK parameter analysis set was subset of safety analysis set (participants who received at least 1 dose of study drug) with participants who had at least 1 of PK parameters of interest for measured analytes related to study drug. Here, ''Number of Participants Analyzed" signifies participants evaluable for this outcome measure and contributed date to the table. Here, 'Number Analyzed' signifies participants evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg)
Number analyzed (Participants) | 3 | 5
Nanograms per milliliter
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 5
  Cycle 1 Day 1 | 5.094 (NA) — Geometric coefficient of variation could not be calculated as at least 3 values were required and this criterion could not be fulfilled due to lack of available data. | 22.81 (80)
  Cycle 1 Day 8: number analyzed (Participants) | 1 | 3
  Cycle 1 Day 8 | 3.440 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 13.74 (106)
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 4
  Cycle 5 Day 1 |  | 33.79 (73)
  Cycle 5 Day 8: number analyzed (Participants) | 1 | 2
  Cycle 5 Day 8 | 13.10 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 24.85 (NA) — Geometric coefficient of variation could not be calculated as at least 3 values were required and this criterion could not be fulfilled due to lack of available data.

50. Secondary Outcome: Phase 1b of Sub-Study B: Cmax of SEA-TGT
Time Frame: Cycle 1: pre-dose, 168 hours post-dose on Day 1, Cycle 5: pre-dose, 168 hours post-dose on Day 1 (1 cycle= 21 days)
Population: PK parameter analysis set: subset of safety analysis set (participants who received at least 1 dose of study drug) with participants who had at least 1 of PK parameters of interest for measured analytes related to study drug. ''Number of Participants Analyzed'': participants evaluable for this outcome measure. 'Number Analyzed': participants evaluable at specified timepoints. Data for only those participants who received SEA-TGT were planned to be reported for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg)
Number analyzed (Participants) | 5
Nanograms per milliliter
  Cycle 1 | 42550 (109)
  Cycle 5: number analyzed (Participants) | 4
  Cycle 5 | 32660 (17)

51. Secondary Outcome: Phase 2 of Sub-Study B: Cmax of Sasanlimab
Time Frame: Cycle 1: pre-dose, 168 hours post-dose on Day 1, Cycle 5: pre-dose, 168 hours post-dose on Day 1 (1 cycle= 21 days)
Population: PK parameter analysis set was subset of safety analysis set (participants who received at least 1 dose of study drug) with participants who had at least 1 of PK parameters of interest for measured analytes related to study drug. 'Number Analyzed' signifies participants evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
Number analyzed (Participants) | 3 | 2 | 7
Nanograms per milliliter
  Cycle 1 | 11780 (45) | 13810 (NA) — Geometric coefficient of variation could not be calculated as at least 3 values were required and this criterion could not be fulfilled due to lack of available data. | 10350 (45)
  Cycle 5: number analyzed (Participants) | 0 | 1 | 1
  Cycle 5 |  | 43500 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 20600 (NA) — Geometric Coefficient of Variation could not be calculated for single participant.

52. Secondary Outcome: Phase 2 of Sub-Study B: Cmax of Axitinib
Time Frame: as for outcome 49
Population: PK parameter analysis set was subset of safety analysis set (participants who received at least 1 dose of study drug) with participants who had at least 1 of PK parameters of interest for measured analytes related to study drug. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Here, 'Number Analyzed' signifies participants evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
Number analyzed (Participants) | 3 | 2 | 6
Nanograms per milliliter
  Cycle 1 Day 1 | 37.43 (85) | 18.23 (NA) — Geometric coefficient of variation could not be calculated as at least 3 values were required and this criterion could not be fulfilled due to lack of available data. | 11.18 (112)
  Cycle 1 Day 8: number analyzed (Participants) | 1 | 1 | 4
  Cycle 1 Day 8 | 39.50 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 2.360 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 2.708 (132)
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 1 | 1
  Cycle 5 Day 1 |  | 11.10 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 7.710 (NA) — Geometric Coefficient of Variation could not be calculated for single participant.
  Cycle 5 Day 8: number analyzed (Participants) | 0 | 0 | 0

53. Secondary Outcome: Phase 2 of Sub-Study B: Cmax of SEA-TGT
Time Frame: Cycle 1: pre-dose, 168 hours post-dose on Day 1, Cycle 5: pre-dose, 168 hours post-dose on Day 1 (1 cycle= 21 days)
Population: PK parameter analysis set was subset of safety analysis set (participants who received at least 1 dose of study drug) with participants who had at least 1 of PK parameters of interest for measured analytes related to study drug. Here, 'Number Analyzed' signifies participants evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
Number analyzed (Participants) | 3 | 2 | 7
Nanograms per milliliter
  Cycle 1 | 36970 (36) | 35500 (NA) — Geometric coefficient of variation could not be calculated as at least 3 values were required and this criterion could not be fulfilled due to lack of available data. | 30590 (39)
  Cycle 5: number analyzed (Participants) | 0 | 1 | 1
  Cycle 5 |  | 43000 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 44900 (NA) — Geometric Coefficient of Variation could not be calculated for single participant.

54. Secondary Outcome: Phase 1b of Sub-Study B: Pre-dose Concentration During Multiple Dosing (Ctrough) of Sasanlimab
Time Frame: Pre-dose on Cycle 1 Day 1 and Cycle 5 Day 1 (1 cycle= 21 days)
Population: PK parameter analysis set was subset of safety analysis set (participants who received at least 1 dose of study drug) with participants who had at least 1 of PK parameters of interest for measured analytes related to study drug. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg)
Number analyzed (Participants) | 2 | 4
Nanograms per milliliter
  Cycle 1: number analyzed (Participants) | 0 | 0
  Cycle 5 | 23000 (NA) — Geometric coefficient of variation could not be calculated as at least 3 values were required and this criterion could not be fulfilled due to lack of available data. | 23170 (29)

55. Secondary Outcome: Phase 1b of Sub-Study B: Pre-dose Concentration During Multiple Dosing (Ctrough) of Axitinib
Time Frame: Pre-dose on Cycle 1 Day 1 and Day 8; pre-dose on Cycle 5 Day 1 and Day 8 (1 cycle= 21 days)
Population: as for outcome 52
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg)
Number analyzed (Participants) | 1 | 3
Nanograms per milliliter
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0
  Cycle 1 Day 8 | 3.440 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 13.74 (106)
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 2
  Cycle 5 Day 1 |  | 29.42 (NA) — Geometric coefficient of variation could not be calculated as at least 3 values were required and this criterion could not be fulfilled due to lack of available data.
  Cycle 5 Day 8: number analyzed (Participants) | 1 | 2
  Cycle 5 Day 8 | 13.10 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 24.85 (NA) — Geometric coefficient of variation could not be calculated as at least 3 values were required and this criterion could not be fulfilled due to lack of available data.

56. Secondary Outcome: Phase 1b of Sub-Study B: Pre-dose Concentration During Multiple Dosing (Ctrough) of SEA-TGT
Time Frame: Pre-dose on Cycle 1 Day 1; pre-dose on Cycle 5 Day 1 (1 cycle= 21 days)
Population: PK parameter analysis set: subset of safety analysis set (participants who received at least 1 dose of study drug) with participants who had at least 1 of PK parameters measured. 'Number of Participants Analyzed': participants evaluable for this outcome measure, 'Number Analyzed': participants evaluable at specified timepoints. Data for only those participants who received SEA-TGT were planned to be reported hence Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) arm was not reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg)
Number analyzed (Participants) | 4
Nanograms per milliliter
  Cycle 1: number analyzed (Participants) | 0
  Cycle 5 | 4813 (35)

57. Secondary Outcome: Phase 2 of Sub-Study B: Pre-dose Concentration During Multiple Dosing (Ctrough) of Sasanlimab
Time Frame: Cycle 1: pre-dose on Day 1, Cycle 5: pre-dose on Day 1 (1 cycle= 21 days)
Population: PK parameter analysis set: subset of safety analysis set (participants who received at least 1 dose of study drug) with participants who had at least 1 of PK parameters of interest for measured analytes related to study drug. 'Number of Participants Analyzed': participants with evaluable data for this outcome measure and 'Number Analyzed': participants evaluable at specified time points. This outcome measure was not applicable for participants of ''Phase 2 of SSB: 1L NSCLC / PD-L1: TPS 1-49%''
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
Number analyzed (Participants) | 0 | 1 | 2
Nanograms per milliliter
  Cycle 1: number analyzed (Participants) | 0 | 0 | 2
  Cycle 1 |  |  | 87.01 (NA) — Geometric coefficient of variation could not be calculated as at least 3 values were required and this criterion could not be fulfilled due to lack of available data.
  Cycle 5: number analyzed (Participants) | 0 | 1 | 1
  Cycle 5 |  | 30400 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 20000 (NA) — Geometric Coefficient of Variation could not be calculated for single participant.

58. Secondary Outcome: Phase 2 of Sub-Study B: Pre-dose Concentration During Multiple Dosing (Ctrough) of Axitinib
Time Frame: Pre-dose on Cycle 1 Day 1 and Day 8; pre-dose on Cycle 5 Day 1 and Day 8 (1 cycle= 21 days)
Population: as for outcome 54
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
Number analyzed (Participants) | 1 | 1 | 4
Nanograms per milliliter
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0
  Cycle 1 Day 8 | 39.50 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 2.360 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 2.708 (132)
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Cycle 5 Day 1 |  |  | 3.630 (NA) — Geometric Coefficient of Variation could not be calculated for single participant.
  Cycle 5 Day 8: number analyzed (Participants) | 0 | 0 | 0

59. Secondary Outcome: Phase 2 of Sub-Study B: Pre-dose Concentration During Multiple Dosing (Ctrough) of SEA-TGT
Time Frame: Pre-dose on Cycle 1 Day 1; pre-dose on Cycle 5 Day 1 (1 cycle= 21 days)
Population: PK parameter analysis set: subset of safety analysis set (participants who received at least 1 dose of study drug) with participants who had at least 1 of PK parameters of interest for measured analytes related to study drug. Here 'Number of Participants Analyzed': participants evaluable for this outcome measure and 'Number Analyzed': participants evaluable at specified time points. This outcome measure was not applicable for participants of ''Phase 2 of SSB: 1L NSCLC / PD-L1: TPS 1-49%''
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
Number analyzed (Participants) | 0 | 1 | 2
Nanograms per milliliter
  Cycle 1 |  | 55.00 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 24.47 (NA) — Geometric coefficient of variation could not be calculated as at least 3 values were required and this criterion could not be fulfilled due to lack of available data.
  Cycle 5: number analyzed (Participants) | 0 | 1 | 1
  Cycle 5 |  | 5770 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 8490 (NA) — Geometric Coefficient of Variation could not be calculated for single participant.

60. Secondary Outcome: Phase 1b of Sub-Study B: Number of Participants With Positive Anti-Drug Antibody (ADA) Against Sasanlimab and SEA-TGT
Description: A participant was considered ADA (or NAb) positive if (1) baseline titer was missing or negative and participant had >= 1 post-treatment positive titer (treatment-induced), or (2) positive titer at baseline and had a >= [4-fold dilution increase] in titer (equivalent to 0.602 unit increase in logarithm to base 10 (log10) titer from baseline in >= 1 post-treatment sample (treatment-boosted).
Time Frame: Pre-dose on Cycle 1 Day 1 until end of treatment (up to approximately 21 months) (1 cycle= 21 days)
Population: Immunogenicity analysis set included participants who had at least 1 analyzed sasanlimab ADA/NAb sample. Here ''Number analyzed'' signifies number of participants with at least one post-treatment ADA result for respective category.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg)
Number analyzed (Participants) | 3 | 6
Participants
  ADA against sasanlimab | 0 | 1
  ADA against SEA-TGT: number analyzed (Participants) | 0 | 6
  ADA against SEA-TGT |  | 0

61. Secondary Outcome: Phase 2 of Sub-Study B: Number of Participants With Positive Anti-Drug Antibody (ADA) Against Sasanlimab and SEA-TGT
Time Frame: Pre-dose on Cycle 1 Day 1 until end of treatment (up to approximately 21 months) (1 cycle= 21 days)
Population: Immunogenicity analysis set included participants who had at least 1 analyzed sasanlimab ADA/NAb sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
Number analyzed (Participants) | 3 | 2 | 7
Participants
  ADA against sasanlimab | 0 | 0 | 0
  ADA against SEA-TGT | 1 | 0 | 0

62. Secondary Outcome: Phase 2 of Sub-Study B: Objective Response Rate by PD-L1 Expression in Available Tumor Tissue
Description: ORR was defined as percentage of participants with confirmed CR or PR according to RECIST v1.1 based on investigator assessment, from the date of first CR or PR until the date of the first documentation of disease progression (PD), death, or start of new anticancer therapy. CR was defined as complete disappearance of all target lesions with exception of nodal disease. All target nodes must decrease to normal size (short axis <10 millimeter [mm]). PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. PD was defined as 20% increase in sum of diameters of target measurable lesions above smallest sum observed (over baseline if no decrease in the sum was observed during therapy), with a minimum absolute increase of 5 mm.
Time Frame: as for outcome 4
Population: Full analysis set included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
Number analyzed (Participants) | 3 | 2 | 7
Percentage of participants | 33.3 [0.8 to 90.6] | 0 [0.0 to 84.2] | 14.3 [0.4 to 57.9]

ADVERSE EVENTS:
Time Frame: From the start of study treatment (Cycle1 Day1) up to 30 days after last dose of study treatment (maximum exposure = 38.66 months; maximum follow-up approximately 39.66 months)
Description: Same event may appear as both non-serious adverse event (non-SAE) and SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. Safety analysis set included all participants who received at least 1 dose of study drug.
Arm/Group | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg) | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg) | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg)
All-Cause Mortality (participants affected / at risk) | 0/4 | 4/9 | 1/3 | 5/6 | 1/3 | 0/2 | 3/7
Serious Adverse Events (participants affected / at risk) | 2/4 | 7/9 | 1/3 | 3/6 | 1/3 | 0/2 | 4/7
Other Adverse Events (participants affected / at risk) | 4/4 | 9/9 | 3/3 | 6/6 | 3/3 | 2/2 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) (N=4) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg) (N=9) | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) (N=3) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg) (N=6) | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) (N=3) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) (N=2) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) (N=7)
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (300mg) + Binimetinib (45mg) (N=4) | Phase 1b of SSA: Sasanlimab (300mg) + Encorafenib (450mg) + Binimetinib (45mg) (N=9) | Phase 1b of SSB: Sasanlimab (225 mg) + Axitinib (5 mg) (N=3) | Phase 1b of SSB: Sasanlimab (225mg) + Axitinib (5 mg) + SEA-TGT(1mg/kg) (N=6) | Phase 2 of SSB: 1L NSCLC PD-L1: TPS 1-49% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) (N=3) | Phase 2 of SSB: 1L NSCLC / PD-L1: TPS >=50% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) (N=2) | Phase 2 of SSB: 2/3L NSCLC / PD-L1: TPS >=1% (Sasanlimab (225mg)+Axitinib (5mg)+SEA-TGT (1mg/kg) (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 2 | 2 | 2 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1
Macular oedema (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Ocular discomfort (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Retinal fovea disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 0 | 2 | 2 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 1 | 3 | 2 | 0 | 3
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 0 | 1 | 2 | 0 | 3
Chest pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 4 | 2 | 3 | 2 | 1 | 3
Oedema peripheral (General disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 1
Acne pustular (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 1 | 2 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 4 | 2 | 1 | 1 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 3 | 1 | 1 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 1 | 1 | 2 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 4 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 2 | 2 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 2 | 0 | 2 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 1 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2 | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 1 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0 | 2 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 2 | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 2 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 4 | 2 | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin tightness (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 3 | 1 | 1 | 1
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 1 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Visceral venous thrombosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site hypersensitivity (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 2 | 1
Amylase increased (Investigations) | 0 | 1 | 0 | 2 | 1 | 0 | 1
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Blood corticotrophin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 2 | 1 | 1 | 0/6
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 1 | 0 | 1 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 2 | 2 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 2 | 3 | 0 | 0 | 2
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Granuloma annulare (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Narrow anterior chamber angle (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nodule (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nodular rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth discolouration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to a business decision, no participant was enrolled in Phase 2 of sub-study A. Hence, Phase 2 was not initiated, and no data was collected and there are no results for this in the record.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from the study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT04585815/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT04585815/SAP_001.pdf